CLINICAL TRIAL: NCT00427908
Title: Evaluate Non-Inferiority and Persistence of the Immune Response of GSK Biologicals' Meningococcal Vaccine 134612 Versus Meningitec™ or Mencevax™ ACWY in Healthy Subjects (1-10 Years of Age)
Brief Title: Study in Children to Evaluate Non-Inferiority and Persistence up to 5 Years of GSK Bio Meningococcal Vaccine 134612
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108658; 108660 (Y1) (Other: GSK); 108661 (Y2) (Other: GSK); 108663 (Y3) (Other: GSK); 108665 (Y4) (Other: GSK); 108668 (Y5) (Other: GSK)
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal serogroups A, C, W-135 and/or Y diseases; Conjugate vaccine; Immunogenicity; Meningococcal vaccine; Persistence; Non-inferiority
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Group A (Experimental): All subjects received GSK Biolgicals' meningococcal vaccine 134612.
  Interventions: Biological: GSK Biolgicals' meningococcal vaccine 134612 (Nimenrix)
- Group B (Active Comparator): Subjects including and above two years of age received Mencevax™ ACWY, subjects below two years of age received Meningitec™.
  Interventions: Biological: Mencevax™ ACWY; Biological: Meningitec™

INTERVENTIONS:
Biological: GSK Biolgicals' meningococcal vaccine 134612 (Nimenrix) — One intramuscular dose.
  Arms: Group A
Biological: Mencevax™ ACWY — One subcutaneous dose.
  Arms: Group B
Biological: Meningitec™ — One intramuscular dose.
  Arms: Group B

SUMMARY:
This study has 2 phases, a vaccination phase and a long-term follow-up phase. In the vaccination phase of this study, the new meningococcal vaccine 134612 will be evaluated in children using Mencevax™ ACWY (in children above 2 years) or Meningitec™ (in children below 2 years) as controls. In the long-term follow-up phase of the study, the long-term protection offered by the vaccines will be assessed up to 5 years after vaccination.

Subjects will be randomized in the primary vaccination phase of the study; no new subjects will be enrolled during the long-term follow-up phase of the study.

DETAILED DESCRIPTION:
Subjects will be enrolled in 3 age strata. Subjects including and above two years of age will receive either GSK Biologicals meningococcal vaccine 134612 or Mencevax™ ACWY, subjects below two years of age will receive either GSK Biologicals meningococcal vaccine 134612 or Meningitec™. All subjects will have 7 blood samples taken: prior and one month after vaccination and one, two, three, four and five years after vaccination.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent or guardian can and will comply with the requirements of the protocol.
* A male or female between, and including, 1 through 10 years of age at the time of vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her parents/guardians' knowledge.

Exclusion Criteria:

For the primary phase:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine(s).
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W, and/or Y (for subjects below 6 years) or within the last five previous years (for subjects 6 years old or above).
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroup A, C, W, and/or Y.
* Previous vaccination with tetanus toxoid containing vaccine within the last 28 days.
* History of meningococcal disease due to serogroup A, C, W, or Y.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

For the long term persistence phase:

* History of meningococcal serogroup A, C, W, and/or Y disease.
* Administration of a meningococcal polysaccharide or a meningococcal polysaccharide conjugate vaccine not planned in the protocol.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 613 (Actual)
Dates: Start 2007-02-07 (Actual); Primary Completion 2007-12-03 (Actual); Study Completion 2007-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Vesikari T, Forsten A, Boutriau D, Bianco V, Van der Wielen M, Miller JM. A randomized study to assess the immunogenicity, antibody persistence and safety of a tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine in children aged 2-10 years. Hum Vaccin Immunother. 2012 Dec 1;8(12):1882-91. doi: 10.4161/hv.22165. Epub 2012 Oct 2. PMID 23032168
- [Background] Vesikari T, Forsten A, Boutriau D, Bianco V, Van der Wielen M, Miller JM. Randomized trial to assess the immunogenicity, safety and antibody persistence up to three years after a single dose of a tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine in toddlers. Hum Vaccin Immunother. 2012 Dec 1;8(12):1892-903. doi: 10.4161/hv.22166. Epub 2012 Oct 2. PMID 23032159
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study is summarised with long term immunogenicity studies 108660 (year 1), 108661 (year 2), 108663 (year 3) and 108665 (year 4) on the GSK Cli

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix 1-2 Years of Age Group: Subjects from 1 to 2 years of age who received one dose of Nimenrix™ vaccine administrated intramuscularly (IM) by injection in the non-dominant deltoid or the thigh region.
- Nimenrix 2-11 Years of Age Group: Subjects from 2 to 11 years of age who received one dose of Nimenrix™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
- Meningitec 1-2 Years of Age Group: Subjects from 1 to 2 years of age who received one dose of Meningitec™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
- Mencevax 2-11 Years of Age Group: Subjects from 2 to 11 years of age who received one dose Mencevax™ vaccine administrated subcutaneous by injection in the non-dominant upper arm.
Period: Primary Phase
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
Started | 229 | 231 | 75 | 78
Completed | 224 | 228 | 72 | 78
Not Completed | 5 | 3 | 3 | 0
Not completed — Lost to Follow-up | 4 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Persistence Phase Year 1
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
Started | 222 | 221 | 71 | 78
Completed | 222 | 221 | 71 | 78
Not Completed | 0 | 0 | 0 | 0
Period: Persistence Phase Year 2
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
Started | 208 | 215 | 53 | 61
Completed | 208 | 215 | 53 | 61
Not Completed | 0 | 0 | 0 | 0
Period: Persistence Phase Year 3
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
Started | 185 | 201 | 38 | 38
Completed | 185 | 201 | 38 | 38
Not Completed | 0 | 0 | 0 | 0
Period: Persistence Phase Year 4
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
Started | 165 | 192 | 34 | 32
Completed | 165 | 192 | 34 | 32
Not Completed | 0 | 0 | 0 | 0
Period: Persistence Phase Year 5
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
Started | 52 | 99 | 12 | 13
Completed | 52 | 99 | 12 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group | Total
Number analyzed (Participants) | 229 | 231 | 75 | 78 | 613
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.1 (2.96) | 71.9 (31.19) | 19.3 (3.07) | 71.8 (30.90) | 45.73 (34.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 115 | 39 | 37 | 307
  Male | 113 | 116 | 36 | 41 | 306
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 0 | 1 | 0 | 0 | 1
  Geographic ancestry: Asian-East Asian heritage | 0 | 1 | 0 | 0 | 1
  Geographic ancestry: White-Arabic/North African heritage | 2 | 1 | 0 | 0 | 3
  Geographic ancestry: White-Caucasian/European heritage | 224 | 225 | 74 | 76 | 599
  Geographic ancestry: Unspecified | 3 | 3 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitides Serogroups A, C, W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Antibodies Vaccine Response
Description: Vaccine response was defined as:
  * for initially seronegative subjects, post vaccination rSBA titer ≥ 1:32
  * for initially seropositive subjects, at least 4-fold increase in rSBA titer from pre to post vaccination.
Time Frame: One Month after vaccination
Population: The analysis was performed on subjects of 2 years and above from the According-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 2-11 Years of Age Primary Phase Group; Mencevax 2-11 Years of Age Primary Phase Group: Pooled group of subjects above 2 years of age, participating in the Primary Phase.
Arm/Group | Nimenrix 2-11 Years of Age Primary Phase Group | Mencevax 2-11 Years of Age Primary Phase Group
Number analyzed (Participants) | 219 | 70
Participants
  rSBA-MenA: number analyzed (Participants) | 185 | 62
  rSBA-MenA | 182 | 57
  rSBA-MenC: number analyzed (Participants) | 212 | 69
  rSBA-MenC | 200 | 56
  rSBA-MenW-135: number analyzed (Participants) | 199 | 68
  rSBA-MenW-135 | 199 | 65
  rSBA-MenY | 217 | 58
Statistical Analysis 1: Comparison: Nimenrix 2-11 Years of Age Primary Phase Group vs Mencevax 2-11 Years of Age Primary Phase Group; To evaluate the non-inferiority of Nimenrix™ conjugate vaccine compared to Mencevax™ plain polysaccharide vaccine in terms of the vaccine response (VRR) to MenA. Response to a vaccine antigen component was defined as: For initially seronegative subject, post-vaccination serum bactericidal assay using rabbit complement (rSBA) titer ≥ 1:32. For initially seropositive subject, at least 4-fold increase in rSBA-MenA titer from pre to post vaccination; Test type: Non-Inferiority — Criterion indicative of non-inferiority: lower limit of the standardized asymptotic 95% confidence interval (CI) for the group difference (Nimenrix minus Mencevax) in the percentage of subjects with bactericidal vaccine response to be greater than or equal to -15% for rSBA-MenA; Difference in percentage = 6.44, 95% CI 2-sided [1.15 to 16.04]
Statistical Analysis 2: Comparison: Nimenrix 2-11 Years of Age Primary Phase Group vs Mencevax 2-11 Years of Age Primary Phase Group; To evaluate the non-inferiority of Nimenrix™ conjugate vaccine compared to Mencevax™ plain polysaccharide vaccine in terms of the vaccine response (VRR) to MenC. Response to a vaccine antigen component was defined as: For initially seronegative subject, post-vaccination serum bactericidal assay using rabbit complement (rSBA) titer ≥ 1:32. For initially seropositive subject, at least 4-fold increase in rSBA-MenC titer from pre to post vaccination; Test type: Non-Inferiority — Criterion indicative of non-inferiority: lower limit of the standardized asymptotic 95% confidence interval (CI) for the group difference (Nimenrix minus Mencevax) in the percentage of subjects with bactericidal vaccine response is greater than or equal to -15% for rSBA-MenC; Difference in percentage = 13.18, 95% CI 2-sided [4.79 to 24.32]
Statistical Analysis 3: Comparison: Nimenrix 2-11 Years of Age Primary Phase Group vs Mencevax 2-11 Years of Age Primary Phase Group; To evaluate the non-inferiority of Nimenrix™ conjugate vaccine compared to Mencevax™ plain polysaccharide vaccine in terms of the vaccine response (VRR) to MenW-135. Response to a vaccine antigen component was defined as: For initially seronegative subject, post-vaccination serum bactericidal assay using rabbit complement (rSBA) titer ≥ 1:32. For initially seropositive subject, at least 4-fold increase in rSBA-MenW-135 titer from pre to post vaccination; Test type: Non-Inferiority — Criterion indicative of non-inferiority: lower limit of the standardized asymptotic 95% confidence interval (CI) for the group difference (Nimenrix minus Mencevax) in the percentage of subjects with bactericidal vaccine response is greater than or equal to -15% for rSBA-MenW-135; Difference in percentage = 4.41, 95% CI 2-sided [1.51 to 12.21]
Statistical Analysis 4: Comparison: Nimenrix 2-11 Years of Age Primary Phase Group vs Mencevax 2-11 Years of Age Primary Phase Group; To evaluate the non-inferiority of Nimenrix™ conjugate vaccine compared to Mencevax™ plain polysaccharide vaccine in terms of the vaccine response (VRR) to MenY. Response to a vaccine antigen component was defined as: For initially seronegative subject, post-vaccination serum bactericidal assay using rabbit complement (rSBA) titer ≥ 1:32. For initially seropositive subject, at least 4-fold increase in rSBA-MenY titer from pre to post vaccination; Test type: Non-Inferiority — Criterion indicative of non-inferiority: lower limit of the standardized asymptotic 95% confidence interval (CI) for the group difference (Nimenrux minus Mencevax) in the percentage of subjects with bactericidal vaccine response is greater than or equal to -15% for rSBA-MenY; Difference in percentage = 16.23, 95% CI 2-sided [8.99 to 26.78]

2. Primary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8. This analysis was performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE) vaccination
Population: The analysis was performed on subjects from 1 to 2 years of age from the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 208 | 67
Participants
  rSBA-MenA: number analyzed (Participants) | 191 | 65
  rSBA-MenA | 81 | 26
  rSBA-MenC: number analyzed (Participants) | 203 | 61
  rSBA-MenC | 80 | 19
  rSBA-MenW-135: number analyzed (Participants) | 208 | 62
  rSBA-MenW-135 | 59 | 24
  rSBA-MenY | 115 | 41

3. Primary Outcome: Percentage of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE) to vaccination
Population: The analysis was performed on subjects of 1 to 2 years of age from the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 208 | 67
Percentage
  rSBA-MenA: number analyzed (Participants) | 191 | 65
  rSBA-MenA | 42.4 [35.3 to 49.8] | 40.0 [28.0 to 52.9]
  rSBA-MenC: number analyzed (Participants) | 203 | 61
  rSBA-MenC | 39.4 [32.6 to 46.5] | 31.1 [19.9 to 44.3]
  rSBA-MenW-135: number analyzed (Participants) | 208 | 62
  rSBA-MenW-135 | 28.4 [22.3 to 35] | 38.7 [26.6 to 51.9]
  rSBA-MenY | 55.3 [48.3 to 62.2] | 61.2 [48.5 to 72.9]

4. Primary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: One month after vaccination [PI(M1)]
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 222 | 68
Participants
  rSBA-MenA: number analyzed (Participants) | 222 | 63
  rSBA-MenA | 222 | 22
  rSBA-MenC: number analyzed (Participants) | 220 | 68
  rSBA-MenC | 220 | 67
  rSBA-MenW-135: number analyzed (Participants) | 222 | 63
  rSBA-MenW-135 | 222 | 27
  rSBA-MenY: number analyzed (Participants) | 222 | 66
  rSBA-MenY | 222 | 49
Statistical Analysis 1: Comparison: Nimenrix 1-2 Years of Age Group vs Meningitec 1-2 Years of Age Group; To evaluate the non-inferiority of the vaccine response induced by Nimenrix™ conjugate vaccine when compared to the licensed Meningitec™ vaccine for MenC as measured by rSBA; Test type: Non-Inferiority — Criterion indicative of non-inferiority (serogroup C only): one month after vaccination, the lower limit of the 2-sided standardized asymptotic 95% CI for the group difference (Nimenrix Group minus Meningitec Group) in the percentage of subjects with rSBA titer ≥ 1:8 is greater than or equal to the predefined clinical limit of -15%; Difference in vaccine response rate = 1.47, 95% CI 2-sided [-0.27 to 7.89]

5. Primary Outcome: Percentage of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: One month after vaccination [PI(M1)]
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 222 | 68
Percentage
  rSBA-MenA: number analyzed (Participants) | 222 | 63
  rSBA-MenA | 100 [98.4 to 100] | 34.9 [23.3 to 48.0]
  rSBA-MenC: number analyzed (Participants) | 220 | 68
  rSBA-MenC | 100 [98.3 to 100] | 98.5 [92.1 to 100]
  rSBA-MenW-135: number analyzed (Participants) | 222 | 63
  rSBA-MenW-135 | 100 [98.4 to 100] | 42.9 [30.5 to 56.0]
  rSBA-MenY: number analyzed (Participants) | 222 | 66
  rSBA-MenY | 100 [98.4 to 100] | 74.2 [62.0 to 84.2]

6. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:128. This analysis was performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Meningitec 1- 2 Years of Age Group: Subjects from 1 to 2 years of age who received one dose of Meningitec™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 222 | 68
Participants
  rSBA-MenA, PRE: number analyzed (Participants) | 191 | 65
  rSBA-MenA, PRE | 59 | 20
  rSBA-MenA, PI(M1): number analyzed (Participants) | 222 | 63
  rSBA-MenA, PI(M1) | 222 | 16
  rSBA-MenC, PRE: number analyzed (Participants) | 203 | 61
  rSBA-MenC, PRE | 29 | 4
  rSBA-MenC, PI(M1): number analyzed (Participants) | 220 | 68
  rSBA-MenC, PI(M1) | 218 | 56
  rSBA-MenW-135, PRE: number analyzed (Participants) | 208 | 62
  rSBA-MenW-135, PRE | 38 | 16
  rSBA-MenW-135, PI(M1): number analyzed (Participants) | 222 | 63
  rSBA-MenW-135, PI(M1) | 222 | 18
  rSBA-MenY, PRE: number analyzed (Participants) | 208 | 67
  rSBA-MenY, PRE | 77 | 28
  rSBA-MenY, PI(M1): number analyzed (Participants) | 222 | 66
  rSBA-MenY, PI(M1) | 221 | 31

7. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs). This analysis was performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 222 | 68
Titers
  rSBA-MenA, PRE: number analyzed (Participants) | 191 | 65
  rSBA-MenA, PRE | 21.6 [16.1 to 29] | 20.2 [12.1 to 33.8]
  rSBA-MenA, PI(M1): number analyzed (Participants) | 222 | 63
  rSBA-MenA, PI(M1) | 3706.5 [3327.2 to 4128.9] | 17.1 [10.1 to 29]
  rSBA-MenC, PRE: number analyzed (Participants) | 203 | 61
  rSBA-MenC, PRE | 13.9 [11 to 17.5] | 9.7 [6.8 to 13.9]
  rSBA-MenC, PI(M1): number analyzed (Participants) | 220 | 68
  rSBA-MenC, PI(M1) | 878.7 [779.4 to 990.7] | 415 [296.9 to 580]
  rSBA-MenW-135, PRE: number analyzed (Participants) | 208 | 62
  rSBA-MenW-135, PRE | 11.3 [8.9 to 14.3] | 16.5 [10.2 to 26.7]
  rSBA-MenW-135, PI(M1): number analyzed (Participants) | 222 | 63
  rSBA-MenW-135, PI(M1) | 5394.6 [4869.9 to 5975.7] | 20.3 [12.5 to 33.2]
  rSBA-MenY, PRE: number analyzed (Participants) | 208 | 67
  rSBA-MenY, PRE | 33.8 [25.6 to 44.6] | 45.3 [27 to 75.8]
  rSBA-MenY, PI(M1): number analyzed (Participants) | 222 | 66
  rSBA-MenY, PI(M1) | 2823.8 [2529 to 3153.1] | 77.1 [46.3 to 128.2]

8. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Values
Description: The cut-off value for the rSBA titers were greater than or equal to ≥ 1:8 and ≥ 1:128. These analyses were performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: The analysis was performed on subjects of 2 years and above from the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2-11 Years of Age Primary Phase Group | Mencevax 2-11 Years of Age Primary Phase Group
Number analyzed (Participants) | 225 | 75
Participants
  rSBA-MenA (PRE) ≥ 1:8: number analyzed (Participants) | 185 | 62
  rSBA-MenA (PRE) ≥ 1:8 | 124 | 40
  rSBA-MenA (PRE) ≥ 1:128: number analyzed (Participants) | 185 | 62
  rSBA-MenA (PRE) ≥ 1:128 | 96 | 32
  rSBA-MenA (PI[M1]) ≥ 1:8 | 225 | 75
  rSBA-MenA (PI[M1]) ≥ 1:128 | 224 | 75
  rSBA-MenC (PRE) ≥ 1:8: number analyzed (Participants) | 212 | 70
  rSBA-MenC (PRE) ≥ 1:8 | 133 | 36
  rSBA-MenC (PRE) ≥ 1:128: number analyzed (Participants) | 212 | 70
  rSBA-MenC (PRE) ≥ 1:128 | 59 | 19
  rSBA-MenC (PI[M1]) ≥ 1:8: number analyzed (Participants) | 225 | 74
  rSBA-MenC (PI[M1]) ≥ 1:8 | 225 | 74
  rSBA-MenC (PI[M1]) ≥ 1:128: number analyzed (Participants) | 225 | 74
  rSBA-MenC (PI[M1]) ≥ 1:128 | 224 | 70
  rSBA-MenW-135 (PRE) ≥ 1:8: number analyzed (Participants) | 199 | 68
  rSBA-MenW-135 (PRE) ≥ 1:8 | 120 | 39
  rSBA-MenW-135 (PRE) ≥ 1:128: number analyzed (Participants) | 199 | 68
  rSBA-MenW-135 (PRE) ≥ 1:128 | 90 | 24
  rSBA-MenW-135 (PI[M1]) ≥ 1:8 | 225 | 75
  rSBA-MenW-135 (PI[M1]) ≥ 1:128 | 225 | 75
  rSBA-MenY (PRE) ≥ 1:8: number analyzed (Participants) | 219 | 70
  rSBA-MenY (PRE) ≥ 1:8 | 147 | 42
  rSBA-MenY (PRE) ≥ 1:128: number analyzed (Participants) | 219 | 70
  rSBA-MenY (PRE) ≥ 1:128 | 98 | 28
  rSBA-MenY (PI[M1]) ≥ 1:8 | 225 | 75
  rSBA-MenY (PI[M1]) ≥ 1:128 | 224 | 73

9. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 7
Time Frame: Prior to (PRE) and one month post vaccination [PI(M1)]
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix 2-11 Years of Age Primary Phase Group | Mencevax 2-11 Years of Age Primary Phase Group
Number analyzed (Participants) | 225 | 75
Titer
  rSBA-MenA (PRE): number analyzed (Participants) | 185 | 62
  rSBA-MenA (PRE) | 57.9 [43.3 to 77.5] | 58.2 [33.8 to 100.1]
  rSBA-MenA (PI[M1]) | 7300.9 [6586 to 8093.4] | 2033.4 [1667.1 to 2480.2]
  rSBA-MenC (PRE): number analyzed (Participants) | 212 | 70
  rSBA-MenC (PRE) | 33.5 [26 to 43.1] | 24.1 [15.2 to 38.2]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 225 | 74
  rSBA-MenC (PI[M1]) | 2435.3 [2105.8 to 2816.3] | 750.2 [555.2 to 1013.7]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 199 | 68
  rSBA-MenW-135 (PRE) | 43.1 [32.4 to 57.4] | 40.1 [23.9 to 67.3]
  rSBA-MenW-135 (PI[M1]) | 11777 [10666.2 to 13003.5] | 2186.3 [1723.1 to 2773.9]
  rSBA-MenY (PRE): number analyzed (Participants) | 219 | 70
  rSBA-MenY (PRE) | 57.3 [43.7 to 75.2] | 45.5 [26.8 to 77]
  rSBA-MenY (PI[M1]) | 6641.4 [6044.3 to 7297.4] | 1409.9 [1085.9 to 1830.5]

10. Secondary Outcome: Number of Subjects With Anti-polysaccharide Meningococcal Serogroup A (Anti-PSA), Serogroup C (Anti-PSC), Serogroup W-135 (Anti-PSW-135) and Serogroup Y (Anti-PSY) Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations were greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL) and ≥ 2.0 μg/mL.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 168 | 51
Participants
  Anti-PSA (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 147 | 43
  Anti-PSA (PRE) ≥ 0.3 μg/mL | 10 | 4
  Anti-PSA (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 147 | 43
  Anti-PSA (PRE) ≥ 2.0 μg/mL | 2 | 1
  Anti-PSA [PI(M1)] ≥ 0.3 μg/mL: number analyzed (Participants) | 162 | 36
  Anti-PSA [PI(M1)] ≥ 0.3 μg/mL | 162 | 2
  Anti-PSA [PI(M1)] ≥ 2.0 μg/mL: number analyzed (Participants) | 162 | 36
  Anti-PSA [PI(M1)] ≥ 2.0 μg/mL | 162 | 1
  Anti-PSC (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 141 | 42
  Anti-PSC (PRE) ≥ 0.3 μg/mL | 3 | 1
  Anti-PSC (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 141 | 42
  Anti-PSC (PRE) ≥ 2.0 μg/mL | 1 | 1
  Anti-PSC [PI(M1)] ≥ 0.3 μg/mL | 168 | 51
  Anti-PSC [PI(M1)] ≥ 2.0 μg/mL | 166 | 50
  Anti-PSW-135 (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 141 | 39
  Anti-PSW-135 (PRE) ≥ 0.3 μg/mL | 2 | 0
  Anti-PSW-135 (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 141 | 39
  Anti-PSW-135 (PRE) ≥ 2.0 μg/mL | 1 | 0
  Anti-PSW-135 [PI(M1)] ≥ 0.3 μg/mL: number analyzed (Participants) | 143 | 36
  Anti-PSW-135 [PI(M1)] ≥ 0.3 μg/mL | 143 | 0
  Anti-PSW-135 [PI(M1)] ≥ 2.0 μg/mL: number analyzed (Participants) | 143 | 36
  Anti-PSW-135 [PI(M1)] ≥ 2.0 μg/mL | 131 | 0
  Anti-PSY (PRE) ≥ 0.3 μg/mL: number analyzed (Participants) | 107 | 30
  Anti-PSY (PRE) ≥ 0.3 μg/mL | 1 | 1
  Anti-PSY (PRE) ≥ 2.0 μg/mL: number analyzed (Participants) | 107 | 30
  Anti-PSY (PRE) ≥ 2.0 μg/mL | 0 | 0
  Anti-PSY [PI(M1)] ≥ 0.3 μg/mL: number analyzed (Participants) | 152 | 32
  Anti-PSY [PI(M1)] ≥ 0.3 μg/mL | 152 | 0
  Anti-PSY [PI(M1)] ≥ 2.0 μg/mL: number analyzed (Participants) | 152 | 32
  Anti-PSY [PI(M1)] ≥ 2.0 μg/mL | 147 | 0

11. Secondary Outcome: Anti-PS Antibody Concentrations
Description: Antibody concentrations are presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 168 | 51
μg/mL
  Anti-PSA (PRE): number analyzed (Participants) | 147 | 43
  Anti-PSA (PRE) | 0.17 [0.15 to 0.18] | 0.18 [0.14 to 0.23]
  Anti-PSA [PI(M1)]: number analyzed (Participants) | 162 | 36
  Anti-PSA [PI(M1)] | 33.36 [29.07 to 38.27] | 0.17 [0.14 to 0.2]
  Anti-PSC (PRE): number analyzed (Participants) | 141 | 42
  Anti-PSC (PRE) | 0.16 [0.15 to 0.17] | 0.16 [0.14 to 0.18]
  Anti-PSC [PI(M1)] | 13.47 [12 to 15.12] | 8.29 [6.8 to 10.1]
  Anti-PSW-135 (PRE): number analyzed (Participants) | 141 | 39
  Anti-PSW-135 (PRE) | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 [PI(M1)]: number analyzed (Participants) | 143 | 36
  Anti-PSW-135 [PI(M1)] | 6.86 [5.87 to 8.02] | 0.15 [0.15 to 0.15]
  Anti-PSY (PRE): number analyzed (Participants) | 107 | 30
  Anti-PSY (PRE) | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.17]
  Anti-PSY [PI(M1)]: number analyzed (Participants) | 152 | 32
  Anti-PSY [PI(M1)] | 10.35 [9.12 to 11.74] | 0.15 [0.15 to 0.15]

12. Secondary Outcome: Number of Subjects With Anti-PS Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations were greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL) and (≥) 2.0 μg/mL.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 2- 11 Years of Age Primary Phase Group; Mencevax 2- 11 Years of Age Primary Phase Group: Pooled group of subjects above 2 years of age, participating in the Primary Phase.
Arm/Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 225 | 75
Participants
  Anti-PSA ≥0.3μg/mL, PRE: number analyzed (Participants) | 218 | 75
  Anti-PSA ≥0.3μg/mL, PRE | 29 | 12
  Anti-PSA ≥0.3μg/mL, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSA ≥0.3μg/mL, PI(M1) | 224 | 73
  Anti-PSA ≥2.0μg/mL, PRE: number analyzed (Participants) | 218 | 75
  Anti-PSA ≥2.0μg/mL, PRE | 9 | 2
  Anti-PSA ≥2.0μg/mL, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSA ≥2.0μg/mL, PI(M1) | 224 | 68
  Anti-PSC ≥0.3μg/mL , PRE: number analyzed (Participants) | 225 | 74
  Anti-PSC ≥0.3μg/mL , PRE | 28 | 6
  Anti-PSC ≥0.3μg/mL, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSC ≥0.3μg/mL, PI(M1) | 224 | 74
  Anti-PSC ≥2.0μg/mL, PRE: number analyzed (Participants) | 225 | 74
  Anti-PSC ≥2.0μg/mL, PRE | 9 | 2
  Anti-PSC ≥2.0μg/mL, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSC ≥2.0μg/mL, PI(M1) | 223 | 71
  Anti-PSW-135 ≥0.3μg/mL, PRE | 3 | 1
  Anti-PSW-135 ≥0.3μg/mL, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSW-135 ≥0.3μg/mL, PI(M1) | 224 | 72
  Anti-PSW-135 ≥2.0μg/mL, PRE | 0 | 0
  Anti-PSW-135 ≥2.0μg/mL, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSW-135 ≥2.0μg/mL, PI(M1) | 197 | 54
  Anti-PSY ≥0.3μg/mL, PRE: number analyzed (Participants) | 224 | 74
  Anti-PSY ≥0.3μg/mL, PRE | 6 | 0
  Anti-PSY ≥0.3μg/mL, PI(M1): number analyzed (Participants) | 225 | 74
  Anti-PSY ≥0.3μg/mL, PI(M1) | 225 | 72
  Anti-PSY ≥2.0μg/mL, PRE: number analyzed (Participants) | 224 | 74
  Anti-PSY ≥2.0μg/mL, PRE | 1 | 0
  Anti-PSY ≥2.0μg/mL, PI(M1): number analyzed (Participants) | 225 | 74
  Anti-PSY ≥2.0μg/mL, PI(M1) | 217 | 71

13. Secondary Outcome: Anti-PS Antibody Concentrations
Description: Antibody concentrations were presented as micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE) and one month post vaccination [PI(M1)]
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 225 | 75
μg/mL
  Anti-PSA, PRE: number analyzed (Participants) | 218 | 75
  Anti-PSA, PRE | 0.19 [0.17 to 0.21] | 0.2 [0.16 to 0.23]
  Anti-PSA, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSA, PI(M1) | 36.35 [32.3 to 40.91] | 10.34 [7.79 to 13.72]
  Anti-PSC, PRE: number analyzed (Participants) | 225 | 74
  Anti-PSC, PRE | 0.2 [0.18 to 0.22] | 0.19 [0.15 to 0.22]
  Anti-PSC, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSC, PI(M1) | 13.33 [11.75 to 15.12] | 14.53 [11.13 to 18.95]
  Anti-PSW-135, PRE | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.16]
  Anti-PSW-135, PI(M1): number analyzed (Participants) | 224 | 74
  Anti-PSW-135, PI(M1) | 6.35 [5.53 to 7.29] | 4.62 [3.37 to 6.35]
  Anti-PSY, PRE: number analyzed (Participants) | 224 | 74
  Anti-PSY, PRE | 0.16 [0.15 to 0.16] | 0.15 [0.15 to 0.15]
  Anti-PSY, PI(M1): number analyzed (Participants) | 225 | 74
  Anti-PSY, PI(M1) | 11.35 [10.01 to 12.87] | 15.45 [11.42 to 20.91]

14. Secondary Outcome: Number of Subjects With Anti-tetanus (Anti-TT) Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-TT concentrations was greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 30 | 6
Participants
  Anti-TT (PRE): number analyzed (Participants) | 19 | 6
  Anti-TT (PRE) | 18 | 5
  Anti-TT [PI(M1)]: number analyzed (Participants) | 30 | 4
  Anti-TT [PI(M1)] | 30 | 4

15. Secondary Outcome: Anti-TT Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs) expressed in international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 30 | 6
IU/mL
  Anti-TT (PRE): number analyzed (Participants) | 19 | 6
  Anti-TT (PRE) | 1.226 [0.609 to 2.47] | 0.57 [0.102 to 3.188]
  Anti-TT [PI(M1)]: number analyzed (Participants) | 30 | 4
  Anti-TT [PI(M1)] | 14.199 [9.628 to 20.94] | 1.341 [0.316 to 5.686]

16. Secondary Outcome: Number of Subjects With Anti-TT Antibody Concentrations
Description: Cut-off values assessed were greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 32 | 7
Participants
  Anti-TT, PRE: number analyzed (Participants) | 19 | 4
  Anti-TT, PRE | 19 | 4
  Anti-TT, PI(M1) | 32 | 7

17. Secondary Outcome: Anti-TT Antibody Concentrations
Description: as for outcome 15
Time Frame: Prior to (PRE) and one month post vaccination [PI(M1)]
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 32 | 7
IU/mL
  Anti-TT, PRE: number analyzed (Participants) | 19 | 4
  Anti-TT, PRE | 1.541 [0.856 to 2.775] | 2.103 [0.129 to 34.398]
  Anti-TT, PI(M1) | 20.951 [14.656 to 29.949] | 1.74 [0.536 to 5.642]

18. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using Human Complement Against Neisseria Meningitides Serogroups A, C, W-135, Y (hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY) Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 221 | 68
Participants
  hSBA-MenA, PRE: number analyzed (Participants) | 215 | 68
  hSBA-MenA, PRE | 3 | 3
  hBA-MenA, PI(M1): number analyzed (Participants) | 217 | 65
  hBA-MenA, PI(M1) | 203 | 4
  hSBA-MenC, PRE: number analyzed (Participants) | 214 | 67
  hSBA-MenC, PRE | 3 | 1
  hSBA-MenC, PI(M1) | 219 | 49
  hSBA-MenW-135, PRE: number analyzed (Participants) | 205 | 64
  hSBA-MenW-135, PRE | 2 | 3
  hSBA-MenW-135, PI(M1): number analyzed (Participants) | 177 | 58
  hSBA-MenW-135, PI(M1) | 145 | 1
  hSBA-MenY, PRE: number analyzed (Participants) | 189 | 57
  hSBA-MenY, PRE | 7 | 2
  hSBA-MenY, PI(M1): number analyzed (Participants) | 201 | 59
  hSBA-MenY, PI(M1) | 135 | 3

19. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 221 | 68
Titers
  hSBA-MenA, PRE: number analyzed (Participants) | 215 | 68
  hSBA-MenA, PRE | 2 [2 to 2.1] | 2.2 [2 to 2.3]
  hBA-MenA, PI(M1): number analyzed (Participants) | 217 | 65
  hBA-MenA, PI(M1) | 59 [49.3 to 70.6] | 2.3 [2 to 2.6]
  hSBA-MenC, PRE: number analyzed (Participants) | 214 | 67
  hSBA-MenC, PRE | 2.1 [2 to 2.2] | 2.1 [1.9 to 2.3]
  hSBA-MenC, PI(M1) | 190 [164.7 to 219.2] | 21.2 [13.9 to 32.3]
  hSBA-MenW-135, PRE: number analyzed (Participants) | 205 | 64
  hSBA-MenW-135, PRE | 2.1 [2 to 2.1] | 2.2 [2 to 2.4]
  hSBA-MenW-135, PI(M1): number analyzed (Participants) | 177 | 58
  hSBA-MenW-135, PI(M1) | 38.8 [29.7 to 50.6] | 2 [2 to 2.1]
  hSBA-MenY, PRE: number analyzed (Participants) | 189 | 57
  hSBA-MenY, PRE | 2.2 [2 to 2.3] | 2.1 [2 to 2.2]
  hSBA-MenY, PI(M1): number analyzed (Participants) | 201 | 59
  hSBA-MenY, PI(M1) | 24.4 [18.6 to 32.1] | 2.4 [1.9 to 3.1]

20. Secondary Outcome: Number of Subjects With hSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: Prior to (PRE) and one month after vaccination [PI(M1)]
Population: The analysis was performed on subjects from 6 to below 11 years of age from the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 6-11 Years of Age Group: Subjects from 6 to 11 years of age who received one dose of Nimenrix™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
- Mencevax 6-11 Years of Age Group: Subjects from 6 to 11 years of age who received one dose Mencevax™ vaccine administrated subcutaneous by injection in the non-dominant upper arm.
Arm/Group | Nimenrix 6-11 Years of Age Group | Mencevax 6-11 Years of Age Group
Number analyzed (Participants) | 112 | 38
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 109 | 36
  hSBA-MenA (PRE) | 2 | 2
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 111 | 35
  hSBA-MenA (PI[M1]) | 91 | 9
  hSBA-MenC (PRE): number analyzed (Participants) | 112 | 35
  hSBA-MenC (PRE) | 35 | 9
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 107 | 38
  hSBA-MenC (PI[M1]) | 96 | 15
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 99 | 30
  hSBA-MenW-135 (PRE) | 13 | 2
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 107 | 35
  hSBA-MenW-135 (PI[M1]) | 102 | 12
  hSBA-MenY (PRE): number analyzed (Participants) | 78 | 24
  hSBA-MenY (PRE) | 24 | 8
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 94 | 32
  hSBA-MenY (PI[M1]) | 79 | 14

21. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE) and one month post vaccination [PI(M1)]
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix 6-11 Years of Age Group | Mencevax 6-11 Years of Age Group
Number analyzed (Participants) | 112 | 38
Titer
  hSBA-MenA (PRE): number analyzed (Participants) | 109 | 36
  hSBA-MenA (PRE) | 2.1 [2.0 to 2.1] | 2.2 [1.9 to 2.5]
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 111 | 35
  hSBA-MenA (PI[M1]) | 57.0 [40.3 to 80.6] | 4.1 [2.6 to 6.5]
  hSBA-MenC (PRE): number analyzed (Participants) | 112 | 35
  hSBA-MenC (PRE) | 5.1 [3.8 to 6.7] | 4.4 [2.7 to 7.2]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 107 | 38
  hSBA-MenC (PI[M1]) | 154.8 [101.1 to 237.1] | 13.1 [5.4 to 32.0]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 99 | 30
  hSBA-MenW-135 (PRE) | 3.2 [2.5 to 4.1] | 2.6 [1.8 to 3.7]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 107 | 35
  hSBA-MenW-135 (PI[M1]) | 134.2 [101.4 to 177.6] | 5.8 [3.3 to 9.9]
  hSBA-MenY (PRE): number analyzed (Participants) | 78 | 24
  hSBA-MenY (PRE) | 5.6 [3.8 to 8.2] | 6.1 [3.0 to 12.6]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 94 | 32
  hSBA-MenY (PI[M1]) | 93.7 [62.1 to 141.4] | 12.5 [5.6 to 27.7]

22. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: The analysis was performed on subjects from 1 to 2 years of age from the ATP cohort for persistence Year 1, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 1 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 216 | 66
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 185 | 64
  rSBA-MenA (PRE) | 80 | 26
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 216 | 61
  rSBA-MenA (PI[M1]) | 216 | 21
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 212 | 49
  rSBA-MenA (PI[M12]) | 210 | 16
  rSBA-MenC (PRE): number analyzed (Participants) | 197 | 61
  rSBA-MenC (PRE) | 78 | 20
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 214 | 66
  rSBA-MenC (PI[M1]) | 214 | 66
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 207 | 63
  rSBA-MenC (PI[M12]) | 203 | 50
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 202 | 62
  rSBA-MenW-135 (PRE) | 57 | 23
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 216 | 61
  rSBA-MenW-135 (PI[M1]) | 216 | 26
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 216 | 64
  rSBA-MenW-135 (PI[M12]) | 216 | 38
  rSBA-MenY (PRE): number analyzed (Participants) | 202 | 66
  rSBA-MenY (PRE) | 113 | 40
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 216 | 65
  rSBA-MenY (PI[M1]) | 216 | 48
  rSBA-MenY (PI[M12]) | 214 | 42

23. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as GMTs. This analysis was performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 216 | 66
Titer
  rSBA-MenA (PRE): number analyzed (Participants) | 185 | 64
  rSBA-MenA (PRE) | 22.6 [16.7 to 30.6] | 20.7 [12.3 to 34.9]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 216 | 61
  rSBA-MenA (PI[M1]) | 3684.2 [3302.8 to 4109.5] | 16.9 [9.9 to 29]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 212 | 49
  rSBA-MenA (PI[M12]) | 967 [843 to 1109.3] | 18.3 [9.5 to 35.1]
  rSBA-MenC (PRE): number analyzed (Participants) | 197 | 61
  rSBA-MenC (PRE) | 14 [11 to 17.6] | 10.2 [7.1 to 14.7]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 214 | 66
  rSBA-MenC (PI[M1]) | 864.2 [763.6 to 978.2] | 448.2 [327.5 to 613.6]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 207 | 63
  rSBA-MenC (PI[M12]) | 195.3 [166.3 to 229.3] | 77.1 [49.1 to 121.1]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 202 | 62
  rSBA-MenW-135 (PRE) | 11.3 [8.9 to 14.4] | 15.5 [9.6 to 24.9]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 216 | 61
  rSBA-MenW-135 (PI[M1]) | 5386.9 [4859.3 to 5971.7] | 20.2 [12.3 to 33.2]
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 216 | 64
  rSBA-MenW-135 (PI[M12]) | 855.1 [757.1 to 965.9] | 36.7 [22.6 to 59.7]
  rSBA-MenY (PRE): number analyzed (Participants) | 202 | 66
  rSBA-MenY (PRE) | 34.6 [26.1 to 45.9] | 44.1 [26.2 to 74.3]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 216 | 65
  rSBA-MenY (PI[M1]) | 2836.5 [2536.4 to 3172] | 78.1 [46.6 to 130.9]
  rSBA-MenY (PI[M12]) | 766.4 [661 to 888.5] | 65.1 [36.9 to 114.7]

24. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: The analysis was performed on subjects of 2 years and above from the ATP cohort for persistence Year 1, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 1 time point.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 2- 11 Years of Age Group: Subjects from 2 to 11 years of age who received one dose of Nimenrix™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
- Mencevax 2- 11 Years of Age Group: Subjects from 2 to 11 years of age who received one dose Mencevax™ vaccine administrated subcutaneous by injection in the non-dominant upper arm.
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 216 | 75
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 175 | 62
  rSBA-MenA (PRE) | 118 | 40
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 214 | 75
  rSBA-MenA (PI[M1]) | 214 | 75
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 216 | 71
  rSBA-MenA (PI[M12]) | 215 | 64
  rSBA-MenC (PRE): number analyzed (Participants) | 202 | 70
  rSBA-MenC (PRE) | 128 | 36
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 214 | 74
  rSBA-MenC (PI[M1]) | 214 | 74
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 215 | 65
  rSBA-MenC (PI[M12]) | 214 | 52
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 190 | 68
  rSBA-MenW-135 (PRE) | 113 | 39
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 214 | 75
  rSBA-MenW-135 (PI[M1]) | 214 | 75
  rSBA-MenW-135 (PI[M12]) | 216 | 75
  rSBA-MenY (PRE): number analyzed (Participants) | 210 | 70
  rSBA-MenY (PRE) | 141 | 42
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 214 | 75
  rSBA-MenY (PI[M1]) | 214 | 75
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 216 | 71
  rSBA-MenY (PI[M12]) | 216 | 64

25. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs). The analysis was performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Mencevax 2- 11 Years of Age Group: Subjects from 2 to 11 years of age who received one dose of Mencevax™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 216 | 75
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 175 | 62
  rSBA-MenA (PRE) | 59.6 [44.1 to 80.3] | 58.2 [33.8 to 100.1]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 214 | 75
  rSBA-MenA (PI[M1]) | 7395.3 [6652.7 to 8220.7] | 2033.4 [1667.1 to 2480.2]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 216 | 71
  rSBA-MenA (PI[M12]) | 2448.1 [2149.6 to 2788.1] | 358.5 [230.2 to 558.4]
  rSBA-MenC (PRE): number analyzed (Participants) | 202 | 70
  rSBA-MenC (PRE) | 34.4 [26.6 to 44.5] | 24.1 [15.2 to 38.2]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 214 | 74
  rSBA-MenC (PI[M1]) | 2488.5 [2145 to 2887] | 750.2 [555.2 to 1013.7]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 215 | 65
  rSBA-MenC (PI[M12]) | 489.5 [419.5 to 571.1] | 113.5 [67.3 to 191.5]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 190 | 68
  rSBA-MenW-135 (PRE) | 41.6 [31.1 to 55.8] | 40.1 [23.9 to 67.3]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 214 | 75
  rSBA-MenW-135 (PI[M1]) | 11943.7 [10782.7 to 13229.7] | 2186.3 [1723.1 to 2773.9]
  rSBA-MenW-135 (PI[M12]) | 2983.3 [2628.2 to 3386.3] | 463 [367.4 to 583.5]
  rSBA-MenY (PRE): number analyzed (Participants) | 210 | 70
  rSBA-MenY (PRE) | 57.4 [43.5 to 75.9] | 45.5 [26.8 to 77]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 214 | 75
  rSBA-MenY (PI[M1]) | 6666.3 [6057.7 to 7336.1] | 1409.9 [1085.9 to 1830.5]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 216 | 71
  rSBA-MenY (PI[M12]) | 2172.1 [1939.6 to 2432.5] | 332.4 [213.5 to 517.7]

26. Secondary Outcome: Number of Subjects With Anti-PS Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 161 | 49
Participants
  Anti-PSA (PRE): number analyzed (Participants) | 142 | 44
  Anti-PSA (PRE) | 9 | 4
  Anti-PSA (PI[M1]): number analyzed (Participants) | 155 | 35
  Anti-PSA (PI[M1]) | 155 | 2
  Anti-PSA (PI[M12]): number analyzed (Participants) | 131 | 38
  Anti-PSA (PI[M12]) | 118 | 3
  Anti-PSC (PRE): number analyzed (Participants) | 137 | 41
  Anti-PSC (PRE) | 3 | 1
  Anti-PSC (PI[M1]) | 161 | 49
  Anti-PSC (PI[M12]): number analyzed (Participants) | 128 | 35
  Anti-PSC (PI[M12]) | 73 | 17
  Anti-PSW-135 (PRE): number analyzed (Participants) | 137 | 38
  Anti-PSW-135 (PRE) | 2 | 0
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 138 | 35
  Anti-PSW-135 (PI[M1]) | 138 | 0
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 132 | 32
  Anti-PSW-135 (PI[M12]) | 124 | 0
  Anti-PSY (PRE): number analyzed (Participants) | 104 | 30
  Anti-PSY (PRE) | 1 | 1
  Anti-PSY (PI[M1]): number analyzed (Participants) | 145 | 31
  Anti-PSY (PI[M1]) | 145 | 0
  Anti-PSY (PI[M12]): number analyzed (Participants) | 157 | 45
  Anti-PSY (PI[M12]) | 153 | 2

27. Secondary Outcome: Anti-PS Antibody Concentrations
Description: Antibody concentrations are presented as GMCs and expressed in micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 161 | 49
μg/mL
  Anti-PSA (PRE): number analyzed (Participants) | 142 | 44
  Anti-PSA (PRE) | 0.17 [0.15 to 0.18] | 0.18 [0.14 to 0.23]
  Anti-PSA (PI[M1]): number analyzed (Participants) | 155 | 35
  Anti-PSA (PI[M1]) | 33.31 [28.94 to 38.35] | 0.17 [0.14 to 0.2]
  Anti-PSA (PI[M12]): number analyzed (Participants) | 131 | 38
  Anti-PSA (PI[M12]) | 1.07 [0.89 to 1.3] | 0.17 [0.15 to 0.18]
  Anti-PSC (PRE): number analyzed (Participants) | 137 | 41
  Anti-PSC (PRE) | 0.16 [0.15 to 0.17] | 0.16 [0.14 to 0.19]
  Anti-PSC (PI[M1]) | 13.44 [11.93 to 15.14] | 8.53 [6.97 to 10.43]
  Anti-PSC (PI[M12]): number analyzed (Participants) | 128 | 35
  Anti-PSC (PI[M12]) | 0.39 [0.33 to 0.46] | 0.34 [0.24 to 0.47]
  Anti-PSW-135 (PRE): number analyzed (Participants) | 137 | 38
  Anti-PSW-135 (PRE) | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 138 | 35
  Anti-PSW-135 (PI[M1]) | 6.87 [5.85 to 8.07] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 132 | 32
  Anti-PSW-135 (PI[M12]) | 1.33 [1.13 to 1.56] | 0.15 [0.15 to 0.15]
  Anti-PSY (PRE): number analyzed (Participants) | 104 | 30
  Anti-PSY (PRE) | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.17]
  Anti-PSY (PI[M1]): number analyzed (Participants) | 145 | 31
  Anti-PSY (PI[M1]) | 10.21 [8.96 to 11.62] | 0.15 [0.15 to 0.15]
  Anti-PSY (PI[M12]): number analyzed (Participants) | 157 | 45
  Anti-PSY (PI[M12]) | 1.97 [1.7 to 2.28] | 0.16 [0.15 to 0.17]

28. Secondary Outcome: Number of Subjects With Anti-PS Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was ≥ 0.3 μg/mL.
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 216 | 75
Participants
  Anti-PSA (PRE): number analyzed (Participants) | 209 | 75
  Anti-PSA (PRE) | 26 | 12
  Anti-PSA (PI[M1]): number analyzed (Participants) | 213 | 74
  Anti-PSA (PI[M1]) | 213 | 73
  Anti-PSA (PI[M12]): number analyzed (Participants) | 213 | 73
  Anti-PSA (PI[M12]) | 209 | 70
  Anti-PSC (PRE): number analyzed (Participants) | 216 | 74
  Anti-PSC (PRE) | 29 | 6
  Anti-PSC (PI[M1]): number analyzed (Participants) | 213 | 74
  Anti-PSC (PI[M1]) | 213 | 74
  Anti-PSC (PI[M12]) | 169 | 74
  Anti-PSW-135 (PRE) | 2 | 1
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 213 | 74
  Anti-PSW-135 (PI[M1]) | 213 | 72
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 210 | 72
  Anti-PSW-135 (PI[M12]) | 206 | 65
  Anti-PSY (PRE): number analyzed (Participants) | 215 | 74
  Anti-PSY (PRE) | 4 | 0
  Anti-PSY (PI[M1]): number analyzed (Participants) | 214 | 74
  Anti-PSY (PI[M1]) | 214 | 72
  Anti-PSY (PI[M12]): number analyzed (Participants) | 215 | 74
  Anti-PSY (PI[M12]) | 213 | 71

29. Secondary Outcome: Anti-PS Antibody Concentrations
Description: Antibody concentrations are presented as GMCs and expressed in μg/mL.
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)] and at Persistence Year 1 [PI(M12)]
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 216 | 75
μg/mL
  Anti-PSA (PRE): number analyzed (Participants) | 209 | 75
  Anti-PSA (PRE) | 0.19 [0.17 to 0.21] | 0.2 [0.16 to 0.23]
  Anti-PSA (PI[M1]): number analyzed (Participants) | 213 | 74
  Anti-PSA (PI[M1]) | 35.95 [31.79 to 40.65] | 10.34 [7.79 to 13.72]
  Anti-PSA (PI[M12]): number analyzed (Participants) | 213 | 73
  Anti-PSA (PI[M12]) | 2.33 [1.94 to 2.79] | 4.05 [2.88 to 5.68]
  Anti-PSC (PRE): number analyzed (Participants) | 216 | 74
  Anti-PSC (PRE) | 0.2 [0.18 to 0.23] | 0.19 [0.15 to 0.22]
  Anti-PSC (PI[M1]): number analyzed (Participants) | 213 | 74
  Anti-PSC (PI[M1]) | 13.34 [11.7 to 15.2] | 14.53 [11.13 to 18.95]
  Anti-PSC (PI[M12]) | 0.76 [0.64 to 0.91] | 4.4 [3.2 to 6.04]
  Anti-PSW-135 (PRE) | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.16]
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 213 | 74
  Anti-PSW-135 (PI[M1]) | 6.26 [5.43 to 7.22] | 4.62 [3.37 to 6.35]
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 210 | 72
  Anti-PSW-135 (PI[M12]) | 1.94 [1.7 to 2.22] | 2.21 [1.54 to 3.15]
  Anti-PSY (PRE): number analyzed (Participants) | 215 | 74
  Anti-PSY (PRE) | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.15]
  Anti-PSY (PI[M1]): number analyzed (Participants) | 214 | 74
  Anti-PSY (PI[M1]) | 11.2 [9.86 to 12.71] | 15.45 [11.42 to 20.91]
  Anti-PSY (PI[M12]): number analyzed (Participants) | 215 | 74
  Anti-PSY (PI[M12]) | 2.76 [2.43 to 3.15] | 5.77 [4.2 to 7.93]

30. Secondary Outcome: Number of Subjects With hSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 215 | 68
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 209 | 66
  hSBA-MenA (PRE) | 3 | 3
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 211 | 63
  hSBA-MenA (PI[M1]) | 196 | 3
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 201 | 63
  hSBA-MenA (PI[M12]) | 47 | 3
  hSBA-MenC (PRE): number analyzed (Participants) | 208 | 65
  hSBA-MenC (PRE) | 3 | 1
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 215 | 66
  hSBA-MenC (PI[M1]) | 213 | 48
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 200 | 64
  hSBA-MenC (PI[M12]) | 192 | 34
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 199 | 62
  hSBA-MenW-135 (PRE) | 2 | 3
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 173 | 56
  hSBA-MenW-135 (PI[M1]) | 141 | 1
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 175 | 62
  hSBA-MenW-135 (PI[M12]) | 172 | 3
  hSBA-MenY (PRE): number analyzed (Participants) | 182 | 55
  hSBA-MenY (PRE) | 7 | 2
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 196 | 57
  hSBA-MenY (PI[M1]) | 131 | 3
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 214 | 68
  hSBA-MenY (PI[M12]) | 200 | 8

31. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 215 | 68
Titers
  hSBA-MenA (PRE): number analyzed (Participants) | 209 | 66
  hSBA-MenA (PRE) | 2 [2 to 2.1] | 2.2 [2 to 2.4]
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 211 | 63
  hSBA-MenA (PI[M1]) | 57.6 [47.9 to 69.3] | 2.2 [1.9 to 2.5]
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 201 | 63
  hSBA-MenA (PI[M12]) | 3.6 [3.1 to 4.2] | 2.2 [2 to 2.4]
  hSBA-MenC (PRE): number analyzed (Participants) | 208 | 65
  hSBA-MenC (PRE) | 2.1 [2 to 2.2] | 2.1 [1.9 to 2.3]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 215 | 66
  hSBA-MenC (PI[M1]) | 187 [161.6 to 216.5] | 22 [14.3 to 33.8]
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 200 | 64
  hSBA-MenC (PI[M12]) | 88.7 [73.8 to 106.5] | 12.2 [7.6 to 19.5]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 199 | 62
  hSBA-MenW-135 (PRE) | 2.1 [2 to 2.2] | 2.2 [2 to 2.4]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 173 | 56
  hSBA-MenW-135 (PI[M1]) | 38.5 [29.3 to 50.5] | 2.1 [2 to 2.2]
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 175 | 62
  hSBA-MenW-135 (PI[M12]) | 225.1 [184.5 to 274.7] | 2.4 [1.9 to 3]
  hSBA-MenY (PRE): number analyzed (Participants) | 182 | 55
  hSBA-MenY (PRE) | 2.2 [2 to 2.3] | 2.1 [2 to 2.2]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 196 | 57
  hSBA-MenY (PI[M1]) | 23.8 [18.1 to 31.4] | 2.5 [1.9 to 3.2]
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 214 | 68
  hSBA-MenY (PI[M12]) | 105.1 [85.2 to 129.7] | 3.2 [2.3 to 4.4]

32. Secondary Outcome: Number of Subjects With hSBA Antibody Titers ≥ to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater or equal to (≥) 1:4.
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)] and Persistence Year 1 [PI(M12)]
Population: The analysis was performed on subjects from 6 to below 11 years of age from the ATP cohort for persistence Year 1, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 1 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 6-11 Years of Age Group | Mencevax 6-11 Years of Age Group
Number analyzed (Participants) | 109 | 38
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 105 | 36
  hSBA-MenA (PRE) | 2 | 2
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 105 | 35
  hSBA-MenA (PI[M1]) | 85 | 9
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 104 | 35
  hSBA-MenA (PI[M12]) | 19 | 4
  hSBA-MenC (PRE]): number analyzed (Participants) | 109 | 35
  hSBA-MenC (PRE]) | 32 | 9
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 101 | 38
  hSBA-MenC (PI[M1]) | 90 | 15
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 105 | 31
  hSBA-MenC (PI[M12]) | 100 | 10
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 95 | 30
  hSBA-MenW-135 (PRE) | 10 | 2
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 103 | 35
  hSBA-MenW-135 (PI[M1]) | 98 | 12
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 103 | 31
  hSBA-MenW-135 (PI[M12]) | 103 | 4
  hSBA-MenY (PRE): number analyzed (Participants) | 75 | 24
  hSBA-MenY (PRE) | 22 | 8
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 89 | 32
  hSBA-MenY (PI[M1]) | 75 | 14
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 106 | 36
  hSBA-MenY (PI[M12]) | 105 | 12

33. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)] and at Persistence Year 1 [PI(M12)]
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix 6-11 Years of Age Group | Mencevax 6-11 Years of Age Group
Number analyzed (Participants) | 109 | 38
Titer
  hSBA-MenA (PRE): number analyzed (Participants) | 105 | 36
  hSBA-MenA (PRE) | 2.1 [2.0 to 2.2] | 2.2 [1.9 to 2.5]
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 105 | 35
  hSBA-MenA (PI[M1]) | 53.4 [37.3 to 76.2] | 4.1 [2.6 to 6.5]
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 104 | 35
  hSBA-MenA (PI[M12]) | 3.5 [2.7 to 4.4] | 2.5 [1.9 to 3.3]
  hSBA-MenC (PRE): number analyzed (Participants) | 109 | 35
  hSBA-MenC (PRE) | 4.7 [3.6 to 6.2] | 4.4 [2.7 to 7.2]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 101 | 38
  hSBA-MenC (PI[M1]) | 155.8 [99.3 to 244.3] | 13.1 [5.4 to 32.0]
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 105 | 31
  hSBA-MenC (PI[M12]) | 129.5 [95.4 to 175.9] | 7.7 [3.5 to 17.3]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 95 | 30
  hSBA-MenW-135 (PRE) | 3.0 [2.3 to 3.8] | 2.6 [1.8 to 3.7]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 103 | 35
  hSBA-MenW-135 (PI[M1]) | 133.5 [99.9 to 178.4] | 5.8 [3.3 to 9.9]
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 103 | 31
  hSBA-MenW-135 (PI[M12]) | 256.7 [218.2 to 301.9] | 3.4 [2.0 to 5.8]
  hSBA-MenY (PRE): number analyzed (Participants) | 75 | 24
  hSBA-MenY (PRE) | 5.3 [3.6 to 7.8] | 6.1 [3.0 to 12.6]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 89 | 32
  hSBA-MenY (PI[M1]) | 95.1 [62.4 to 145.1] | 12.5 [5.6 to 27.7]
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 106 | 36
  hSBA-MenY (PI[M12]) | 265.0 [213.0 to 329.6] | 9.3 [4.3 to 19.9]

34. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: The analysis was performed on subjects from 1 to 2 years of age from the ATP cohort for persistence Year 2, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 2 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 199 | 52
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 171 | 48
  rSBA-MenA (PRE) | 73 | 21
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 199 | 47
  rSBA-MenA (PI[M1]) | 199 | 18
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 195 | 36
  rSBA-MenA (PI[M12]) | 193 | 13
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 190 | 45
  rSBA-MenA (PI[M24]) | 188 | 30
  rSBA-MenC (PRE): number analyzed (Participants) | 181 | 47
  rSBA-MenC (PRE) | 72 | 16
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 197 | 50
  rSBA-MenC (PI[M1]) | 197 | 50
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 189 | 47
  rSBA-MenC (PI[M12]) | 188 | 47
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 197 | 52
  rSBA-MenC (PI[M24]) | 185 | 38
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 188 | 47
  rSBA-MenW-135 (PRE) | 54 | 16
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 199 | 48
  rSBA-MenW-135 (PI[M1]) | 199 | 19
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 198 | 49
  rSBA-MenW-135 (PI[M12]) | 198 | 29
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 199 | 44
  rSBA-MenW-135 (PI[M24]) | 198 | 24
  rSBA-MenY (PRE): number analyzed (Participants) | 185 | 50
  rSBA-MenY (PRE) | 104 | 31
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 199 | 50
  rSBA-MenY (PI[M1]) | 199 | 38
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 198 | 50
  rSBA-MenY (PI[M12]) | 196 | 35
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 197 | 50
  rSBA-MenY (PI[M24]) | 193 | 37

35. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 7
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 199 | 52
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 171 | 48
  rSBA-MenA (PRE) | 22.7 [16.5 to 31.2] | 24 [12.9 to 44.6]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 199 | 47
  rSBA-MenA (PI[M1]) | 3743 [3341.1 to 4193.2] | 20 [10.6 to 37.8]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 195 | 36
  rSBA-MenA (PI[M12]) | 961.4 [830 to 1113.5] | 21.5 [9.8 to 47]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 190 | 45
  rSBA-MenA (PI[M24]) | 567.7 [489.8 to 658] | 51.3 [29 to 90.8]
  rSBA-MenC (PRE): number analyzed (Participants) | 181 | 47
  rSBA-MenC (PRE) | 13.7 [10.8 to 17.5] | 11.2 [7.2 to 17.4]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 197 | 50
  rSBA-MenC (PI[M1]) | 870.9 [766 to 990.1] | 626.4 [442.7 to 886.3]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 189 | 47
  rSBA-MenC (PI[M12]) | 203.9 [174.2 to 238.6] | 163.7 [118.6 to 226]
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 197 | 52
  rSBA-MenC (PI[M24]) | 117.4 [97.1 to 141.9] | 57.7 [33.5 to 99.3]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 188 | 47
  rSBA-MenW-135 (PRE) | 11.5 [8.9 to 14.7] | 13 [7.8 to 21.8]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 199 | 48
  rSBA-MenW-135 (PI[M1]) | 5424.4 [4867.9 to 6044.4] | 17.6 [10.2 to 30.5]
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 198 | 49
  rSBA-MenW-135 (PI[M12]) | 856.6 [755.4 to 971.3] | 35.4 [20.4 to 61.5]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 199 | 44
  rSBA-MenW-135 (PI[M24]) | 415.9 [362.4 to 477.3] | 27.5 [15.7 to 48.1]
  rSBA-MenY (PRE): number analyzed (Participants) | 185 | 50
  rSBA-MenY (PRE) | 34 [25.4 to 45.5] | 44.6 [24.8 to 80.2]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 199 | 50
  rSBA-MenY (PI[M1]) | 2797.6 [2494.9 to 3137.1] | 86 [49.3 to 150]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 198 | 50
  rSBA-MenY (PI[M12]) | 749.4 [642.9 to 873.6] | 82.7 [44.7 to 152.9]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 197 | 50
  rSBA-MenY (PI[M24]) | 504.1 [421 to 603.6] | 93.5 [51.8 to 168.7]

36. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was ≥ 1:8. This analysis was performed by the GSK Biologicals' laboratory.
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: The analysis was performed on subjects of 2 years and above from the ATP cohort for persistence Year 2, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 2 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 210 | 59
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 170 | 48
  rSBA-MenA (PRE) | 113 | 32
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenA (PI[M1]) | 209 | 59
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 208 | 57
  rSBA-MenA (PI[M12]) | 207 | 53
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 208 | 56
  rSBA-MenA (PI[M24]) | 208 | 51
  rSBA-MenC (PRE): number analyzed (Participants) | 196 | 56
  rSBA-MenC (PRE) | 125 | 34
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenC (PI[M1]) | 209 | 59
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 207 | 49
  rSBA-MenC (PI[M12]) | 207 | 49
  rSBA-MenC (PI[M24]) | 207 | 39
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 189 | 53
  rSBA-MenW-135 (PRE) | 115 | 32
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenW-135 (PI[M1]) | 209 | 59
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 208 | 59
  rSBA-MenW-135 (PI[M12]) | 208 | 59
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 210 | 54
  rSBA-MenW-135 (PI[M24]) | 209 | 46
  rSBA-MenY (PRE): number analyzed (Participants) | 204 | 54
  rSBA-MenY (PRE) | 138 | 31
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenY (PI[M1]) | 209 | 59
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 208 | 55
  rSBA-MenY (PI[M12]) | 208 | 52
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 210 | 55
  rSBA-MenY (PI[M24]) | 210 | 41

37. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 7
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 36
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Nimenrix 2- 11 Years of Age Group; Mencevax 2- 11 Years of Age Group: Pooled group of subjects above 2 years of age.
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 210 | 59
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 170 | 48
  rSBA-MenA (PRE) | 57.1 [42.1 to 77.4] | 64.5 [34.9 to 119]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenA (PI[M1]) | 7392.2 [6645 to 8223.3] | 2230.8 [1797.6 to 2768.3]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 208 | 57
  rSBA-MenA (PI[M12]) | 2475.3 [2170.5 to 2822.9] | 450.6 [289 to 702.7]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 208 | 56
  rSBA-MenA (PI[M24]) | 1333.4 [1181.9 to 1504.2] | 202.5 [135.3 to 303]
  rSBA-MenC (PRE): number analyzed (Participants) | 196 | 56
  rSBA-MenC (PRE) | 35.4 [27.2 to 46] | 33.7 [20 to 56.8]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenC (PI[M1]) | 2475.6 [2128.8 to 2878.9] | 966.7 [695.7 to 1343.2]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 207 | 49
  rSBA-MenC (PI[M12]) | 490.3 [421.7 to 570.2] | 277 [187.4 to 409.6]
  rSBA-MenC (PI[M24]) | 256 [213.9 to 306.2] | 59.9 [33 to 108.7]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 189 | 53
  rSBA-MenW-135 (PRE) | 43.9 [32.8 to 58.8] | 46.2 [25.7 to 83]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenW-135 (PI[M1]) | 11892.6 [10744.2 to 13163.7] | 2215 [1679.2 to 2921.7]
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 208 | 59
  rSBA-MenW-135 (PI[M12]) | 2969.7 [2612.5 to 3375.9] | 496.2 [383.5 to 641.9]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 210 | 54
  rSBA-MenW-135 (PI[M24]) | 1298 [1135.5 to 1483.7] | 144 [90.1 to 230.2]
  rSBA-MenY (PRE): number analyzed (Participants) | 204 | 54
  rSBA-MenY (PRE) | 58.3 [44 to 77.3] | 40.9 [22.3 to 75]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 209 | 59
  rSBA-MenY (PI[M1]) | 6594.5 [5971.2 to 7282.9] | 1574.2 [1177.1 to 2105.3]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 208 | 55
  rSBA-MenY (PI[M12]) | 2115.5 [1886.4 to 2372.5] | 418 [269.2 to 649.2]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 210 | 55
  rSBA-MenY (PI[M24]) | 1530.2 [1339.2 to 1748.4] | 96.9 [54.1 to 173.6]

38. Secondary Outcome: Anti-PS Antibody Concentrations
Description: as for outcome 11
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 161 | 39
μg/mL
  Anti-PSA (PRE): number analyzed (Participants) | 132 | 35
  Anti-PSA (PRE) | 0.16 [0.15 to 0.18] | 0.19 [0.14 to 0.25]
  Anti-PSA (PI[M1]): number analyzed (Participants) | 143 | 27
  Anti-PSA (PI[M1]) | 32.63 [28.2 to 37.75] | 0.18 [0.14 to 0.22]
  Anti-PSA (PI[M12]): number analyzed (Participants) | 121 | 31
  Anti-PSA (PI[M12]) | 1.08 [0.89 to 1.32] | 0.16 [0.14 to 0.18]
  Anti-PSA (PI[M24]): number analyzed (Participants) | 140 | 39
  Anti-PSA (PI[M24]) | 0.59 [0.5 to 0.69] | 0.19 [0.16 to 0.23]
  Anti-PSC (PRE): number analyzed (Participants) | 126 | 31
  Anti-PSC (PRE) | 0.16 [0.15 to 0.17] | 0.16 [0.14 to 0.2]
  Anti-PSC (PI[M1]): number analyzed (Participants) | 148 | 35
  Anti-PSC (PI[M1]) | 13.58 [12.01 to 15.36] | 9.16 [7.31 to 11.47]
  Anti-PSC (PI[M12]): number analyzed (Participants) | 117 | 30
  Anti-PSC (PI[M12]) | 0.39 [0.33 to 0.47] | 0.36 [0.24 to 0.53]
  Anti-PSC (PI[M24]): number analyzed (Participants) | 107 | 22
  Anti-PSC (PI[M24]) | 0.26 [0.22 to 0.3] | 0.24 [0.17 to 0.36]
  Anti-PSW-135 (PRE): number analyzed (Participants) | 127 | 29
  Anti-PSW-135 (PRE) | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 129 | 24
  Anti-PSW-135 (PI[M1]) | 6.58 [5.6 to 7.74] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 122 | 26
  Anti-PSW-135 (PI[M12]) | 1.33 [1.12 to 1.58] | 0.15 [0.15 to 0.15]
  Anti-PSW-135 (PI[M24]): number analyzed (Participants) | 135 | 32
  Anti-PSW-135 (PI[M24]) | 0.65 [0.54 to 0.79] | 0.15 [0.15 to 0.15]
  Anti-PSY (PRE): number analyzed (Participants) | 96 | 22
  Anti-PSY (PRE) | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.18]
  Anti-PSY (PI[M1]): number analyzed (Participants) | 135 | 24
  Anti-PSY (PI[M1]) | 10.22 [8.96 to 11.67] | 0.15 [0.15 to 0.15]
  Anti-PSY (PI[M12]): number analyzed (Participants) | 144 | 35
  Anti-PSY (PI[M12]) | 1.95 [1.67 to 2.27] | 0.15 [0.15 to 0.17]
  Anti-PSY (PI[M24]): number analyzed (Participants) | 161 | 33
  Anti-PSY (PI[M24]) | 1.12 [0.96 to 1.3] | 0.16 [0.14 to 0.19]

39. Secondary Outcome: Number of Subjects With Anti-PS Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was ≥ 0.3 micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 161 | 39
Participants
  Anti-PSA (PRE): number analyzed (Participants) | 132 | 35
  Anti-PSA (PRE) | 7 | 4
  Anti-PSA (PI[M1]): number analyzed (Participants) | 143 | 27
  Anti-PSA (PI[M1]) | 143 | 2
  Anti-PSA (PI[M12]): number analyzed (Participants) | 121 | 31
  Anti-PSA (PI[M12]) | 109 | 2
  Anti-PSA (PI[M24]): number analyzed (Participants) | 140 | 39
  Anti-PSA (PI[M24]) | 107 | 7
  Anti-PSC (PRE): number analyzed (Participants) | 126 | 31
  Anti-PSC (PRE) | 3 | 1
  Anti-PSC (PI[M1]): number analyzed (Participants) | 148 | 35
  Anti-PSC (PI[M1]) | 148 | 35
  Anti-PSC (PI[M12]): number analyzed (Participants) | 117 | 30
  Anti-PSC (PI[M12]) | 68 | 15
  Anti-PSC (PI[M24]): number analyzed (Participants) | 107 | 22
  Anti-PSC (PI[M24]) | 38 | 6
  Anti-PSW-135 (PRE): number analyzed (Participants) | 127 | 29
  Anti-PSW-135 (PRE) | 1 | 0
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 129 | 24
  Anti-PSW-135 (PI[M1]) | 129 | 0
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 122 | 26
  Anti-PSW-135 (PI[M12]) | 114 | 0
  Anti-PSW-135 (PI[M24]): number analyzed (Participants) | 135 | 32
  Anti-PSW-135 (PI[M24]) | 98 | 0
  Anti-PSY (PRE): number analyzed (Participants) | 96 | 22
  Anti-PSY (PRE) | 1 | 1
  Anti-PSY (PI[M1]): number analyzed (Participants) | 135 | 24
  Anti-PSY (PI[M1]) | 135 | 0
  Anti-PSY (PI[M12]): number analyzed (Participants) | 144 | 35
  Anti-PSY (PI[M12]) | 140 | 1
  Anti-PSY (PI[M24]): number analyzed (Participants) | 161 | 33
  Anti-PSY (PI[M24]) | 144 | 1

40. Secondary Outcome: Number of Subjects With Anti-PS Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was ≥ 0.3 micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 210 | 59
Participants
  Anti-PSA (PRE): number analyzed (Participants) | 203 | 59
  Anti-PSA (PRE) | 24 | 11
  Anti-PSA (PI[M1]): number analyzed (Participants) | 208 | 59
  Anti-PSA (PI[M1]) | 208 | 58
  Anti-PSA (PI[M12]): number analyzed (Participants) | 205 | 57
  Anti-PSA (PI[M12]) | 201 | 54
  Anti-PSA (PI[M24]): number analyzed (Participants) | 199 | 56
  Anti-PSA (PI[M24]) | 187 | 54
  Anti-PSC (PRE): number analyzed (Participants) | 210 | 58
  Anti-PSC (PRE) | 29 | 6
  Anti-PSC (PI[M1]): number analyzed (Participants) | 208 | 59
  Anti-PSC (PI[M1]) | 208 | 59
  Anti-PSC (PI[M12]): number analyzed (Participants) | 208 | 59
  Anti-PSC (PI[M12]) | 163 | 58
  Anti-PSC (PI[M24]): number analyzed (Participants) | 208 | 59
  Anti-PSC (PI[M24]) | 131 | 57
  Anti-PSW-135 (PRE) | 3 | 1
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 208 | 59
  Anti-PSW-135 (PI[M1]) | 208 | 57
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 202 | 57
  Anti-PSW-135 (PI[M12]) | 198 | 52
  Anti-PSW-135 (PI[M24]): number analyzed (Participants) | 204 | 58
  Anti-PSW-135 (PI[M24]) | 181 | 52
  Anti-PSY (PRE): number analyzed (Participants) | 209 | 58
  Anti-PSY (PRE) | 5 | 0
  Anti-PSY (PI[M1]): number analyzed (Participants) | 209 | 58
  Anti-PSY (PI[M1]) | 209 | 56
  Anti-PSY (PI[M12]): number analyzed (Participants) | 207 | 59
  Anti-PSY (PI[M12]) | 205 | 56
  Anti-PSY (PI[M24]): number analyzed (Participants) | 205 | 54
  Anti-PSY (PI[M24]) | 198 | 50

41. Secondary Outcome: Anti-PS Antibody Concentrations
Description: Antibody concentrations are presented as GMCs and expressed in micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 36
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 210 | 59
μg/mL
  Anti-PSA (PRE): number analyzed (Participants) | 203 | 59
  Anti-PSA (PRE) | 0.18 [0.17 to 0.2] | 0.21 [0.17 to 0.26]
  Anti-PSA (PI[M1]): number analyzed (Participants) | 208 | 59
  Anti-PSA (PI[M1]) | 34.76 [30.83 to 39.19] | 11.2 [8.1 to 15.47]
  Anti-PSA (PI[M12]): number analyzed (Participants) | 205 | 57
  Anti-PSA (PI[M12]) | 2.27 [1.9 to 2.71] | 4.62 [3.13 to 6.82]
  Anti-PSA (PI[M24]): number analyzed (Participants) | 199 | 56
  Anti-PSA (PI[M24]) | 1.52 [1.28 to 1.81] | 2.93 [2.07 to 4.14]
  Anti-PSC (PRE): number analyzed (Participants) | 210 | 58
  Anti-PSC (PRE) | 0.2 [0.18 to 0.23] | 0.2 [0.16 to 0.25]
  Anti-PSC (PI[M1]): number analyzed (Participants) | 208 | 59
  Anti-PSC (PI[M1]) | 12.94 [11.37 to 14.72] | 15.28 [11.24 to 20.77]
  Anti-PSC (PI[M12]): number analyzed (Participants) | 208 | 59
  Anti-PSC (PI[M12]) | 0.75 [0.63 to 0.9] | 4.98 [3.51 to 7.06]
  Anti-PSC (PI[M24]): number analyzed (Participants) | 208 | 59
  Anti-PSC (PI[M24]) | 0.54 [0.45 to 0.64] | 2.81 [2.02 to 3.91]
  Anti-PSW-135 (PRE) | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.16]
  Anti-PSW-135 (PI[M1]): number analyzed (Participants) | 208 | 59
  Anti-PSW-135 (PI[M1]) | 6.16 [5.34 to 7.11] | 4.5 [3.13 to 6.47]
  Anti-PSW-135 (PI[M12]): number analyzed (Participants) | 202 | 57
  Anti-PSW-135 (PI[M12]) | 1.9 [1.66 to 2.17] | 2.28 [1.53 to 3.4]
  Anti-PSW-135 (PI[M24]): number analyzed (Participants) | 204 | 58
  Anti-PSW-135 (PI[M24]) | 1.15 [0.99 to 1.34] | 1.32 [0.92 to 1.9]
  Anti-PSY (PRE): number analyzed (Participants) | 209 | 58
  Anti-PSY (PRE) | 0.16 [0.15 to 0.16] | 0.15 [0.15 to 0.15]
  Anti-PSY (PI[M1]): number analyzed (Participants) | 209 | 58
  Anti-PSY (PI[M1]) | 11.1 [9.76 to 12.63] | 14.91 [10.45 to 21.28]
  Anti-PSY (PI[M12]): number analyzed (Participants) | 207 | 59
  Anti-PSY (PI[M12]) | 2.73 [2.39 to 3.11] | 5.8 [4.01 to 8.39]
  Anti-PSY (PI[M24]): number analyzed (Participants) | 205 | 54
  Anti-PSY (PI[M24]) | 1.72 [1.49 to 1.98] | 2.9 [1.98 to 4.26]

42. Secondary Outcome: Number of Subjects With hSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 198 | 52
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 193 | 51
  hSBA-MenA (PRE) | 3 | 3
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 194 | 48
  hSBA-MenA (PI[M1]) | 180 | 2
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 185 | 47
  hSBA-MenA (PI[M12]) | 42 | 3
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 180 | 50
  hSBA-MenA (PI[M24]) | 73 | 6
  hSBA-MenC (PRE): number analyzed (Participants) | 192 | 49
  hSBA-MenC (PRE) | 2 | 1
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 198 | 50
  hSBA-MenC (PI[M1]) | 196 | 38
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 185 | 50
  hSBA-MenC (PI[M12]) | 179 | 28
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 191 | 51
  hSBA-MenC (PI[M24]) | 179 | 28
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 183 | 47
  hSBA-MenW-135 (PRE) | 2 | 2
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 158 | 45
  hSBA-MenW-135 (PI[M1]) | 130 | 1
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 159 | 46
  hSBA-MenW-135 (PI[M12]) | 156 | 3
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 178 | 51
  hSBA-MenW-135 (PI[M24]) | 171 | 5
  hSBA-MenY (PRE): number analyzed (Participants) | 168 | 42
  hSBA-MenY (PRE) | 6 | 2
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 181 | 44
  hSBA-MenY (PI[M1]) | 121 | 3
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 196 | 52
  hSBA-MenY (PI[M12]) | 183 | 8
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 173 | 43
  hSBA-MenY (PI[M24]) | 157 | 13

43. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)] and Persistence Year 2 [PI(M24)]
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 198 | 52
Titers
  hSBA-MenA (PRE): number analyzed (Participants) | 193 | 51
  hSBA-MenA (PRE) | 2 [2 to 2.1] | 2.2 [2 to 2.5]
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 194 | 48
  hSBA-MenA (PI[M1]) | 58.8 [48.5 to 71.3] | 2.2 [1.9 to 2.7]
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 185 | 47
  hSBA-MenA (PI[M12]) | 3.6 [3.0 to 4.2] | 2.2 [2.0 to 2.6]
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 180 | 50
  hSBA-MenA (PI[M24]) | 5.1 [4.2 to 6.1] | 2.3 [2 to 2.5]
  hSBA-MenC (PRE): number analyzed (Participants) | 192 | 49
  hSBA-MenC (PRE) | 2.1 [2 to 2.1] | 2.1 [1.9 to 2.4]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 198 | 50
  hSBA-MenC (PI[M1]) | 185.4 [159.3 to 215.9] | 26.7 [16.1 to 44.3]
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 185 | 50
  hSBA-MenC (PI[M12]) | 88.6 [73.6 to 106.6] | 14.7 [8.4 to 25.6]
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 191 | 51
  hSBA-MenC (PI[M24]) | 55.6 [45.1 to 68.5] | 11.8 [6.8 to 20.6]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 183 | 47
  hSBA-MenW-135 (PRE) | 2.1 [2 to 2.2] | 2.1 [2 to 2.3]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 158 | 45
  hSBA-MenW-135 (PI[M1]) | 38.7 [29.2 to 51.2] | 2.1 [1.9 to 2.2]
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 159 | 46
  hSBA-MenW-135 (PI[M12]) | 218.8 [177.1 to 270.5] | 2.6 [1.9 to 3.5]
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 178 | 51
  hSBA-MenW-135 (PI[M24]) | 111.4 [90.9 to 136.5] | 2.9 [2.1 to 4]
  hSBA-MenY (PRE): number analyzed (Participants) | 168 | 42
  hSBA-MenY (PRE) | 2.1 [2 to 2.3] | 2.1 [2 to 2.2]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 181 | 44
  hSBA-MenY (PI[M1]) | 23.1 [17.4 to 30.8] | 2.6 [1.9 to 3.7]
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 196 | 52
  hSBA-MenY (PI[M12]) | 99.8 [80.2 to 124.0] | 3.7 [2.4 to 5.6]
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 173 | 43
  hSBA-MenY (PI[M24]) | 72.5 [57 to 92.4] | 5 [3.1 to 7.9]

44. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)] and Persistence Year 3 [PI(M36)]
Population: The analysis was performed on subjects from 1 to 2 years of age from the ATP cohort for persistence Year 3, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 3 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 177 | 37
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 151 | 35
  rSBA-MenA (PRE) | 65 | 15
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 177 | 32
  rSBA-MenA (PI[M1]) | 177 | 10
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 174 | 22
  rSBA-MenA (PI[M12]) | 172 | 7
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 165 | 30
  rSBA-MenA (PI[M24]) | 164 | 21
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 170 | 32
  rSBA-MenA (PI[M36]) | 168 | 27
  rSBA-MenC (PRE): number analyzed (Participants) | 163 | 34
  rSBA-MenC (PRE) | 71 | 12
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 175 | 36
  rSBA-MenC (PI[M1]) | 175 | 36
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 169 | 35
  rSBA-MenC (PI[M12]) | 169 | 35
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 171 | 36
  rSBA-MenC (PI[M24]) | 171 | 36
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 174 | 37
  rSBA-MenC (PI[M36]) | 158 | 36
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 167 | 33
  rSBA-MenW-135 (PRE) | 50 | 11
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 177 | 36
  rSBA-MenW-135 (PI[M1]) | 177 | 14
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 176 | 35
  rSBA-MenW-135 (PI[M12]) | 176 | 22
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 173 | 30
  rSBA-MenW-135 (PI[M24]) | 172 | 15
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 174 | 33
  rSBA-MenW-135 (PI[M36]) | 172 | 24
  rSBA-MenY (PRE): number analyzed (Participants) | 166 | 36
  rSBA-MenY (PRE) | 96 | 24
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 177 | 36
  rSBA-MenY (PI[M1]) | 177 | 29
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 176 | 35
  rSBA-MenY (PI[M12]) | 175 | 24
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 171 | 35
  rSBA-MenY (PI[M24]) | 168 | 27
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 177 | 36
  rSBA-MenY (PI[M36]) | 174 | 33

45. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).This analysis was performed by the GSK Biologicals' laboratory.
Time Frame: as for outcome 44
Population: as for outcome 44
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 177 | 37
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 151 | 35
  rSBA-MenA (PRE) | 23 [16.4 to 32.2] | 21.8 [10.8 to 44.1]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 177 | 32
  rSBA-MenA (PI[M1]) | 3787.4 [3353.2 to 4277.8] | 14.4 [7 to 29.4]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 174 | 22
  rSBA-MenA (PI[M12]) | 974.4 [831 to 1142.4] | 17.6 [6.5 to 47.6]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 165 | 30
  rSBA-MenA (PI[M24]) | 575.2 [494 to 669.9] | 56.5 [28.5 to 112.2]
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 170 | 32
  rSBA-MenA (PI[M36]) | 518.6 [447.6 to 600.8] | 117.1 [65 to 211.2]
  rSBA-MenC (PRE): number analyzed (Participants) | 163 | 34
  rSBA-MenC (PRE) | 15.5 [11.9 to 20] | 12 [6.9 to 20.9]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 175 | 36
  rSBA-MenC (PI[M1]) | 887 [770.4 to 1021.2] | 727.6 [478.7 to 1105.8]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 169 | 35
  rSBA-MenC (PI[M12]) | 223.5 [192.2 to 259.8] | 218.3 [157.9 to 301.8]
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 171 | 36
  rSBA-MenC (PI[M24]) | 141.2 [120.3 to 165.6] | 158.6 [103.8 to 242.2]
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 174 | 37
  rSBA-MenC (PI[M36]) | 125.1 [96.7 to 162] | 185.7 [118.3 to 291.5]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 167 | 33
  rSBA-MenW-135 (PRE) | 11.7 [9 to 15.1] | 12.6 [6.8 to 23.5]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 177 | 36
  rSBA-MenW-135 (PI[M1]) | 5563.5 [4976.9 to 6219.4] | 17.5 [9.2 to 33.6]
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 176 | 35
  rSBA-MenW-135 (PI[M12]) | 904.9 [792.5 to 1033.2] | 37.9 [20.1 to 71.3]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 173 | 30
  rSBA-MenW-135 (PI[M24]) | 439.3 [379 to 509.4] | 22.9 [11.6 to 45.1]
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 174 | 33
  rSBA-MenW-135 (PI[M36]) | 439.8 [370.5 to 522] | 64.5 [33.5 to 124.3]
  rSBA-MenY (PRE): number analyzed (Participants) | 166 | 36
  rSBA-MenY (PRE) | 37.4 [27.4 to 51] | 52.5 [26.7 to 103.3]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 177 | 36
  rSBA-MenY (PI[M1]) | 2875.6 [2540 to 3255.6] | 101.5 [54.3 to 189.7]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 176 | 35
  rSBA-MenY (PI[M12]) | 799.2 [683.3 to 934.7] | 75.7 [36.2 to 158.3]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 171 | 35
  rSBA-MenY (PI[M24]) | 532.8 [439.7 to 645.6] | 100.6 [50.6 to 200]
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 177 | 36
  rSBA-MenY (PI[M36]) | 583.2 [479 to 709.9] | 176 [97.6 to 317.3]

46. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 7
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)] and at Persistence Year 3 [PI(M36)]
Population: The analysis was performed on subjects from of 2 years and above from the ATP cohort for persistence Year 3, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 3 time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 196 | 37
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 162 | 31
  rSBA-MenA (PRE) | 58.4 [42.8 to 79.6] | 69.8 [30.6 to 158.8]
  rSBA-MenA (PI[M1]) | 7513.7 [6740.4 to 8375.7] | 2244.3 [1737.7 to 2898.6]
  rSBA-MenA (PI[M12]) | 2533.4 [2211.6 to 2902.1] | 576.2 [334.8 to 991.7]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 193 | 35
  rSBA-MenA (PI[M24]) | 1352.7 [1191.4 to 1535.7] | 240.1 [149.5 to 385.7]
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 192 | 34
  rSBA-MenA (PI[M36]) | 1184.2 [1054.2 to 1330.3] | 218.8 [128.9 to 371.5]
  rSBA-MenC (PRE): number analyzed (Participants) | 184 | 35
  rSBA-MenC (PRE) | 36.5 [27.8 to 48] | 61.3 [31.4 to 119.7]
  rSBA-MenC (PI[M1]) | 2524.9 [2162.1 to 2948.5] | 1433.7 [939.4 to 2188]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 195 | 34
  rSBA-MenC (PI[M12]) | 509.4 [439.4 to 590.6] | 437.6 [282.9 to 676.8]
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 195 | 37
  rSBA-MenC (PI[M24]) | 273.1 [229.3 to 325.1] | 237.9 [144 to 393]
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 192 | 37
  rSBA-MenC (PI[M36]) | 244.3 [200.8 to 297.3] | 163.5 [83.8 to 319.2]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 173 | 33
  rSBA-MenW-135 (PRE) | 45.4 [33.5 to 61.5] | 57.4 [27.6 to 119.4]
  rSBA-MenW-135 (PI[M1]) | 12158.8 [10949.9 to 13501.1] | 2602.6 [1795.6 to 3772.4]
  rSBA-MenW-135 (PI[M12]) | 3064.7 [2692.8 to 3488] | 587 [411.3 to 837.9]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 195 | 34
  rSBA-MenW-135 (PI[M24]) | 1324.4 [1154.4 to 1519.4] | 182.8 [104 to 321.2]
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 196 | 35
  rSBA-MenW-135 (PI[M36]) | 1737.1 [1503.8 to 2006.7] | 112.9 [59.9 to 212.6]
  rSBA-MenY (PRE): number analyzed (Participants) | 192 | 34
  rSBA-MenY (PRE) | 55.4 [41.3 to 74.3] | 37.2 [17.3 to 80.4]
  rSBA-MenY (PI[M1]) | 6655.7 [6009.1 to 7372] | 1813.8 [1235.6 to 2662.5]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 196 | 34
  rSBA-MenY (PI[M12]) | 2164 [1924.2 to 2433.6] | 467.5 [261.3 to 836.5]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 195 | 37
  rSBA-MenY (PI[M24]) | 1556.4 [1355.9 to 1786.6] | 116.2 [59.3 to 227.7]
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 195 | 37
  rSBA-MenY (PI[M36]) | 1551.6 [1381.2 to 1743.1] | 103.8 [54.3 to 198.3]

47. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)] and Persistence Year 3 [PI(M36)]
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 196 | 37
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 162 | 31
  rSBA-MenA (PRE) | 109 | 20
  rSBA-MenA (PI[M1]) | 196 | 37
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 196 | 36
  rSBA-MenA (PI[M12]) | 195 | 34
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 193 | 35
  rSBA-MenA (PI[M24]) | 193 | 33
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 192 | 34
  rSBA-MenA (PI[M36]) | 192 | 31
  rSBA-MenC (PRE): number analyzed (Participants) | 184 | 35
  rSBA-MenC (PRE) | 118 | 26
  rSBA-MenC (PI[M1]) | 196 | 37
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 195 | 34
  rSBA-MenC (PI[M12]) | 195 | 34
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 195 | 37
  rSBA-MenC (PI[M24]) | 195 | 37
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 192 | 37
  rSBA-MenC (PI[M36]) | 189 | 31
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 173 | 33
  rSBA-MenW-135 (PRE) | 107 | 22
  rSBA-MenW-135 (PI[M1]) | 196 | 37
  rSBA-MenW-135 (PI[M12]) | 196 | 37
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 195 | 34
  rSBA-MenW-135 (PI[M24]) | 194 | 30
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 196 | 35
  rSBA-MenW-135 (PI[M36]) | 196 | 29
  rSBA-MenY (PRE): number analyzed (Participants) | 192 | 34
  rSBA-MenY (PRE) | 127 | 19
  rSBA-MenY (PI[M1]) | 196 | 37
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 196 | 34
  rSBA-MenY (PI[M12]) | 196 | 32
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 195 | 37
  rSBA-MenY (PI[M24]) | 195 | 30
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 195 | 37
  rSBA-MenY (PI[M36]) | 195 | 30

48. Secondary Outcome: Number of Subjects With hSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: as for outcome 47
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 176 | 37
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 172 | 37
  hSBA-MenA (PRE) | 1 | 3
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 172 | 36
  hSBA-MenA (PI[M1]) | 159 | 3
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 163 | 34
  hSBA-MenA (PI[M12]) | 35 | 2
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 157 | 35
  hSBA-MenA (PI[M24]) | 62 | 5
  hSBA-MenA (PI[M36]): number analyzed (Participants) | 170 | 36
  hSBA-MenA (PI[M36]) | 37 | 2
  hSBA-MenC (PRE): number analyzed (Participants) | 170 | 35
  hSBA-MenC (PRE) | 2 | 0
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 176 | 36
  hSBA-MenC (PI[M1]) | 174 | 31
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 162 | 35
  hSBA-MenC (PI[M12]) | 159 | 24
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 165 | 35
  hSBA-MenC (PI[M24]) | 158 | 23
  hSBA-MenC (PI[M36]): number analyzed (Participants) | 166 | 33
  hSBA-MenC (PI[M36]) | 147 | 25
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 163 | 34
  hSBA-MenW-135 (PRE) | 2 | 2
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 138 | 33
  hSBA-MenW-135 (PI[M1]) | 112 | 1
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 143 | 34
  hSBA-MenW-135 (PI[M12]) | 141 | 1
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 153 | 35
  hSBA-MenW-135 (PI[M24]) | 147 | 4
  hSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 164 | 35
  hSBA-MenW-135 (PI[M36]) | 131 | 3
  hSBA-MenY (PRE): number analyzed (Participants) | 149 | 31
  hSBA-MenY (PRE) | 5 | 2
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 161 | 34
  hSBA-MenY (PI[M1]) | 110 | 3
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 174 | 37
  hSBA-MenY (PI[M12]) | 163 | 6
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 149 | 31
  hSBA-MenY (PI[M24]) | 133 | 12
  hSBA-MenY (PI[M36]): number analyzed (Participants) | 159 | 33
  hSBA-MenY (PI[M36]) | 117 | 9

49. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: as for outcome 47
Population: as for outcome 44
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 176 | 37
Titers
  hSBA-MenA (PRE): number analyzed (Participants) | 172 | 37
  hSBA-MenA (PRE) | 2 [2 to 2] | 2.3 [2 to 2.7]
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 172 | 36
  hSBA-MenA (PI[M1]) | 56.9 [46.4 to 69.9] | 2.4 [1.9 to 3]
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 163 | 34
  hSBA-MenA (PI[M12]) | 3.4 [2.9 to 4.1] | 2.2 [1.9 to 2.7]
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 157 | 35
  hSBA-MenA (PI[M24]) | 4.9 [4.0 to 6.0] | 2.3 [2.0 to 2.7]
  hSBA-MenA (PI[M36]): number analyzed (Participants) | 170 | 36
  hSBA-MenA (PI[M36]) | 3.3 [2.8 to 3.8] | 2.2 [1.9 to 2.6]
  hSBA-MenC (PRE): number analyzed (Participants) | 170 | 35
  hSBA-MenC (PRE) | 2.1 [2 to 2.2] | 2 [2 to 2]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 176 | 36
  hSBA-MenC (PI[M1]) | 182.7 [154.6 to 215.8] | 44.1 [25.2 to 77.3]
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 162 | 35
  hSBA-MenC (PI[M12]) | 95.1 [79.1 to 114.5] | 23.8 [12.3 to 46.1]
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 165 | 35
  hSBA-MenC (PI[M24]) | 62.9 [50.9 to 77.8] | 18.8 [9.2 to 38.4]
  hSBA-MenC (PI[M36]): number analyzed (Participants) | 166 | 33
  hSBA-MenC (PI[M36]) | 65.1 [49.6 to 85.5] | 32.5 [16 to 65.9]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 163 | 34
  hSBA-MenW-135 (PRE) | 2.1 [2 to 2.2] | 2.2 [1.9 to 2.6]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 138 | 33
  hSBA-MenW-135 (PI[M1]) | 39.1 [28.8 to 53.1] | 2.1 [1.9 to 2.3]
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 143 | 34
  hSBA-MenW-135 (PI[M12]) | 218.9 [176.3 to 271.9] | 2.1 [1.9 to 2.4]
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 153 | 35
  hSBA-MenW-135 (PI[M24]) | 112.8 [90.6 to 140.4] | 3.1 [2.0 to 4.8]
  hSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 164 | 35
  hSBA-MenW-135 (PI[M36]) | 40.8 [31.1 to 53.6] | 3 [1.9 to 4.7]
  hSBA-MenY (PRE): number analyzed (Participants) | 149 | 31
  hSBA-MenY (PRE) | 2.1 [2 to 2.2] | 2.1 [1.9 to 2.3]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 161 | 34
  hSBA-MenY (PI[M1]) | 24.8 [18.3 to 33.5] | 2.8 [1.8 to 4.4]
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 174 | 37
  hSBA-MenY (PI[M12]) | 103.5 [81.7 to 131.0] | 3.7 [2.3 to 5.9]
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 149 | 31
  hSBA-MenY (PI[M24]) | 70.4 [53.9 to 91.8] | 6.7 [3.7 to 12.3]
  hSBA-MenY (PI[M36]): number analyzed (Participants) | 159 | 33
  hSBA-MenY (PI[M36]) | 37.3 [27.2 to 51.2] | 6 [3 to 11.9]

50. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 2
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)], Persistence Year 3 [PI(M36)] and Persistence Year 4 [PI(M48)]
Population: The analysis was performed on subjects from 1 to 2 years of age from the ATP cohort for persistence Year 4, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 4 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 152 | 31
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 130 | 30
  rSBA-MenA (PRE) | 62 | 11
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 152 | 26
  rSBA-MenA (PI[M1]) | 152 | 7
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 150 | 19
  rSBA-MenA (PI[M12]) | 148 | 6
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 143 | 28
  rSBA-MenA (PI[M24]) | 142 | 19
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 144 | 26
  rSBA-MenA (PI[M36]) | 143 | 22
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 136 | 24
  rSBA-MenA (PI[M48]) | 133 | 21
  rSBA-MenC (PRE): number analyzed (Participants) | 138 | 30
  rSBA-MenC (PRE) | 57 | 13
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 150 | 29
  rSBA-MenC (PI[M1]) | 150 | 29
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 146 | 29
  rSBA-MenC (PI[M12]) | 146 | 29
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 148 | 31
  rSBA-MenC (PI[M24]) | 148 | 31
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 148 | 30
  rSBA-MenC (PI[M36]) | 147 | 30
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 137 | 30
  rSBA-MenC (PI[M48]) | 125 | 27
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 143 | 28
  rSBA-MenW-135 (PRE) | 44 | 8
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 152 | 29
  rSBA-MenW-135 (PI[M1]) | 152 | 12
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 152 | 29
  rSBA-MenW-135 (PI[M12]) | 152 | 17
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 149 | 25
  rSBA-MenW-135 (PI[M24]) | 148 | 12
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 147 | 28
  rSBA-MenW-135 (PI[M36]) | 146 | 20
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 138 | 27
  rSBA-MenW-135 (PI[M48]) | 133 | 18
  rSBA-MenY (PRE): number analyzed (Participants) | 143 | 31
  rSBA-MenY (PRE) | 83 | 21
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 152 | 29
  rSBA-MenY (PI[M1]) | 152 | 25
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 152 | 30
  rSBA-MenY (PI[M12]) | 151 | 22
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 147 | 30
  rSBA-MenY (PI[M24]) | 146 | 23
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 150 | 29
  rSBA-MenY (PI[M36]) | 148 | 27
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 138 | 29
  rSBA-MenY (PI[M48]) | 134 | 23

51. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 7
Time Frame: as for outcome 50
Population: as for outcome 50
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 152 | 31
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 130 | 30
  rSBA-MenA (PRE) | 27.9 [19.2 to 40.4] | 18.1 [8.3 to 39.3]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 152 | 26
  rSBA-MenA (PI[M1]) | 3911.7 [3443.2 to 4444] | 12.4 [5.6 to 27.4]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 150 | 19
  rSBA-MenA (PI[M12]) | 938.4 [790.3 to 1114.3] | 15.9 [5.6 to 45]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 143 | 28
  rSBA-MenA (PI[M24]) | 533 [451.6 to 629] | 53.8 [25.9 to 112]
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 144 | 26
  rSBA-MenA (PI[M36]) | 503 [432.3 to 585.3] | 129.3 [65.9 to 254]
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 136 | 24
  rSBA-MenA (PI[M48]) | 623.9 [507.1 to 767.6] | 157.4 [79.1 to 313]
  rSBA-MenC (PRE): number analyzed (Participants) | 138 | 30
  rSBA-MenC (PRE) | 14.9 [11.2 to 19.9] | 15.4 [8.3 to 28.5]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 150 | 29
  rSBA-MenC (PI[M1]) | 922.5 [794.7 to 1070.8] | 846.2 [537.3 to 1332.8]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 146 | 29
  rSBA-MenC (PI[M12]) | 236.8 [199.7 to 280.7] | 233.9 [160.3 to 341.5]
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 148 | 31
  rSBA-MenC (PI[M24]) | 162.5 [138.2 to 191.1] | 185.3 [116.9 to 293.6]
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 148 | 30
  rSBA-MenC (PI[M36]) | 176.1 [138.6 to 223.9] | 210.3 [139.6 to 316.8]
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 137 | 30
  rSBA-MenC (PI[M48]) | 141.9 [103.8 to 194] | 150.5 [73.4 to 308.6]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 143 | 28
  rSBA-MenW-135 (PRE) | 11.9 [9 to 15.7] | 10.9 [5.6 to 21.3]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 152 | 29
  rSBA-MenW-135 (PI[M1]) | 5495.6 [4864.5 to 6208.6] | 19.8 [9.3 to 41.8]
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 152 | 29
  rSBA-MenW-135 (PI[M12]) | 900.8 [782.6 to 1036.8] | 36.5 [17.5 to 76.1]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 149 | 25
  rSBA-MenW-135 (PI[M24]) | 426.3 [364 to 499.3] | 24.1 [10.8 to 54.1]
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 147 | 28
  rSBA-MenW-135 (PI[M36]) | 454.9 [382.7 to 540.7] | 62.8 [30.4 to 129.5]
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 138 | 27
  rSBA-MenW-135 (PI[M48]) | 400.9 [316.6 to 507.7] | 59.8 [26.5 to 135.1]
  rSBA-MenY (PRE): number analyzed (Participants) | 143 | 31
  rSBA-MenY (PRE) | 37.9 [27.1 to 53.1] | 52.7 [25.7 to 108.3]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 152 | 29
  rSBA-MenY (PI[M1]) | 2839.7 [2497.7 to 3228.4] | 123.9 [66.4 to 231.4]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 152 | 30
  rSBA-MenY (PI[M12]) | 776.5 [655 to 920.5] | 87.8 [40.7 to 189.5]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 147 | 30
  rSBA-MenY (PI[M24]) | 539.2 [444.7 to 653.7] | 100 [47 to 212.5]
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 150 | 29
  rSBA-MenY (PI[M36]) | 581.5 [472.5 to 715.6] | 220.9 [117.8 to 414.2]
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 138 | 29
  rSBA-MenY (PI[M48]) | 524.2 [417 to 658.9] | 174.1 [74.6 to 406.6]

52. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: as for outcome 2
Time Frame: as for outcome 50
Population: The analysis was performed on subjects of 2 years and above from the ATP cohort for persistence Year 4, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 4 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 188 | 29
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 155 | 24
  rSBA-MenA (PRE) | 105 | 14
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenA (PI[M1]) | 187 | 29
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 188 | 28
  rSBA-MenA (PI[M12]) | 188 | 26
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 185 | 27
  rSBA-MenA (PI[M24]) | 185 | 25
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 182 | 27
  rSBA-MenA (PI[M36]) | 182 | 24
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 188 | 28
  rSBA-MenA (PI[M48]) | 188 | 24
  rSBA-MenC (PRE): number analyzed (Participants) | 176 | 28
  rSBA-MenC (PRE) | 112 | 22
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenC (PI[M1]) | 187 | 29
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 187 | 28
  rSBA-MenC (PI[M12]) | 187 | 28
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 186 | 29
  rSBA-MenC (PI[M24]) | 186 | 29
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 181 | 29
  rSBA-MenC (PI[M36]) | 181 | 27
  rSBA-MenC (PI[M48]) | 182 | 26
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 165 | 27
  rSBA-MenW-135 (PRE) | 104 | 19
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenW-135 (PI[M1]) | 187 | 29
  rSBA-MenW-135 (PI[M12]) | 188 | 29
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 186 | 26
  rSBA-MenW-135 (PI[M24]) | 185 | 22
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 185 | 28
  rSBA-MenW-135 (PI[M36]) | 185 | 22
  rSBA-MenW-135 (PI[M48]) | 188 | 22
  rSBA-MenY (PRE): number analyzed (Participants) | 183 | 26
  rSBA-MenY (PRE) | 123 | 14
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenY (PI[M1]) | 187 | 29
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 188 | 27
  rSBA-MenY (PI[M12]) | 188 | 26
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 186 | 29
  rSBA-MenY (PI[M24]) | 186 | 23
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 185 | 29
  rSBA-MenY (PI[M36]) | 185 | 24
  rSBA-MenY (PI[M48]) | 188 | 24

53. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 7
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)], Persistence Year 3 [PI(M36)] and Persistence Year 4 [PI(M48)]
Population: as for outcome 52
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 188 | 29
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 155 | 24
  rSBA-MenA (PRE) | 59.5 [43.4 to 81.7] | 58.3 [21.1 to 160.9]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenA (PI[M1]) | 7593.9 [6848.5 to 8420.4] | 2075.1 [1544.1 to 2788.7]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 188 | 28
  rSBA-MenA (PI[M12]) | 2556.2 [2260.3 to 2890.9] | 488.7 [246.6 to 968.3]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 185 | 27
  rSBA-MenA (PI[M24]) | 1317.2 [1155.9 to 1500.9] | 203.2 [112.6 to 366.5]
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 182 | 27
  rSBA-MenA (PI[M36]) | 1154.1 [1026.8 to 1297.2] | 193.8 [102.1 to 367.9]
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 188 | 28
  rSBA-MenA (PI[M48]) | 1932.3 [1684.9 to 2216.1] | 182.8 [85.5 to 390.9]
  rSBA-MenC (PRE): number analyzed (Participants) | 176 | 28
  rSBA-MenC (PRE) | 35.8 [27 to 47.4] | 69.7 [34 to 142.9]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenC (PI[M1]) | 2578.5 [2221.9 to 2992.3] | 1371.7 [837.1 to 2247.7]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 187 | 28
  rSBA-MenC (PI[M12]) | 510.1 [439.3 to 592.4] | 444.8 [271.1 to 729.9]
  rSBA-MenC (PI[M24]): number analyzed (Participants) | 186 | 29
  rSBA-MenC (PI[M24]) | 278.5 [234.3 to 330.9] | 307.4 [179.2 to 527.4]
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 181 | 29
  rSBA-MenC (PI[M36]) | 255.7 [211.3 to 309.4] | 260 [136.9 to 493.8]
  rSBA-MenC (PI[M48]) | 203.6 [162.9 to 254.6] | 211.9 [104.8 to 428.7]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 165 | 27
  rSBA-MenW-135 (PRE) | 47.4 [34.8 to 64.6] | 63.7 [28.7 to 141.5]
  rSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenW-135 (PI[M1]) | 12275.6 [11099.2 to 13576.7] | 2428 [1565 to 3767.1]
  rSBA-MenW-135 (PI[M12]) | 3083.8 [2712.1 to 3506.3] | 564.2 [366 to 869.7]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 186 | 26
  rSBA-MenW-135 (PI[M24]) | 1324.2 [1150.3 to 1524.3] | 149.4 [72.4 to 308.1]
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 185 | 28
  rSBA-MenW-135 (PI[M36]) | 1748.3 [1508.7 to 2025.9] | 95.7 [44.5 to 205.8]
  rSBA-MenW-135 (PI[M48]) | 1807.5 [1568.9 to 2082.5] | 93.4 [44.2 to 197.5]
  rSBA-MenY (PRE): number analyzed (Participants) | 183 | 26
  rSBA-MenY (PRE) | 56.8 [42.2 to 76.6] | 34.7 [14 to 86]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 187 | 29
  rSBA-MenY (PI[M1]) | 6801.4 [6206.1 to 7453.9] | 1696.6 [1103.1 to 2609.4]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 188 | 27
  rSBA-MenY (PI[M12]) | 2169.8 [1930.4 to 2438.9] | 480.4 [260.9 to 884.9]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 186 | 29
  rSBA-MenY (PI[M24]) | 1550.8 [1352.6 to 1778] | 106.6 [48.5 to 234.1]
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 185 | 29
  rSBA-MenY (PI[M36]) | 1551.5 [1378.9 to 1745.7] | 101.6 [50 to 206.5]
  rSBA-MenY (PI[M48]) | 1545.5 [1356.6 to 1760.6] | 113.1 [55.1 to 232.3]

54. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs). This analysis was performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Persistence Year 4 [PI(M48)]
Population: as for outcome 50
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 152 | 31
Titers
  rSBA-MenA (PI[M48]) | 25.7 [19.1 to 34.7] | 4 [4 to 4]
  rSBA-MenC (PI[M48]) | 11.2 [8.3 to 15.1] | 11.4 [5.2 to 25]
  rSBA-MenW-135 (PI[M48]) | 31.3 [21.4 to 45.6] | 4 [4 to 4]
  rSBA-MenY (PI[M48]) | 29.9 [21.5 to 41.6] | 12.5 [6 to 26.1]

55. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8. This analysis was performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Persistence Year 4 [PI(M48)]
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 152 | 31
Participants
  rSBA-MenA (PI[M48]) | 93 | 0
  rSBA-MenC (PI[M48]) | 46 | 8
  rSBA-MenW-135 (PI[M48]) | 78 | 0
  rSBA-MenY (PI[M48]) | 84 | 9

56. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: as for outcome 55
Time Frame: At Persistence Year 4 [PI(M48)]
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 188 | 29
Participants
  rSBA-MenA (PI[M48]) | 157 | 5
  rSBA-MenC (PI[M48]) | 94 | 12
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 187 | 29
  rSBA-MenW-135 (PI[M48]) | 169 | 4
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 187 | 29
  rSBA-MenY (PI[M48]) | 151 | 2

57. Secondary Outcome: rSBA Antibody Titers (HPA Laboratory Assay)
Description: as for outcome 54
Time Frame: At Persistence Year 4 [PI(M48)]
Population: as for outcome 52
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 188 | 29
Titers
  rSBA-MenA (PI[M48]) | 77.5 [59.3 to 101.3] | 7.3 [4.3 to 12.4]
  rSBA-MenC (PI[M48]) | 21.7 [16.2 to 29.1] | 23.5 [9.8 to 56.3]
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 187 | 29
  rSBA-MenW-135 (PI[M48]) | 671.1 [500.8 to 899.4] | 7.6 [4 to 14.4]
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 187 | 29
  rSBA-MenY (PI[M48]) | 134.8 [99.1 to 183.5] | 4.7 [3.5 to 6.4]

58. Secondary Outcome: Number of Subjects With hSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)], Persistence Year 3 [PI(M36)], Persistence Year 4 [PI(M48)]
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 151 | 31
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 148 | 30
  hSBA-MenA (PRE) | 0 | 2
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 148 | 30
  hSBA-MenA (PI[M1]) | 137 | 1
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 140 | 28
  hSBA-MenA (PI[M12]) | 29 | 1
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 137 | 30
  hSBA-MenA (PI[M24]) | 53 | 4
  hSBA-MenA (PI[M36]): number analyzed (Participants) | 143 | 29
  hSBA-MenA (PI[M36]) | 32 | 1
  hSBA-MenA (PI[M48]): number analyzed (Participants) | 140 | 31
  hSBA-MenA (PI[M48]) | 57 | 8
  hSBA-MenC (PRE): number analyzed (Participants) | 146 | 28
  hSBA-MenC (PRE) | 2 | 0
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 151 | 29
  hSBA-MenC (PI[M1]) | 149 | 25
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 139 | 30
  hSBA-MenC (PI[M12]) | 135 | 22
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 142 | 30
  hSBA-MenC (PI[M24]) | 135 | 22
  hSBA-MenC (PI[M36]): number analyzed (Participants) | 140 | 26
  hSBA-MenC (PI[M36]) | 129 | 21
  hSBA-MenC (PI[M48]): number analyzed (Participants) | 147 | 31
  hSBA-MenC (PI[M48]) | 126 | 24
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 141 | 27
  hSBA-MenW-135 (PRE) | 2 | 1
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 119 | 28
  hSBA-MenW-135 (PI[M1]) | 100 | 1
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 121 | 28
  hSBA-MenW-135 (PI[M12]) | 118 | 1
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 134 | 30
  hSBA-MenW-135 (PI[M24]) | 129 | 5
  hSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 139 | 28
  hSBA-MenW-135 (PI[M36]) | 114 | 2
  hSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 143 | 31
  hSBA-MenW-135 (PI[M48]) | 117 | 3
  hSBA-MenY (PRE): number analyzed (Participants) | 127 | 26
  hSBA-MenY (PRE) | 5 | 1
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 139 | 28
  hSBA-MenY (PI[M1]) | 93 | 2
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 150 | 31
  hSBA-MenY (PI[M12]) | 141 | 5
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 132 | 26
  hSBA-MenY (PI[M24]) | 119 | 10
  hSBA-MenY (PI[M36]): number analyzed (Participants) | 133 | 27
  hSBA-MenY (PI[M36]) | 102 | 7
  hSBA-MenY (PI[M48]): number analyzed (Participants) | 129 | 26
  hSBA-MenY (PI[M48]) | 100 | 12

59. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: as for outcome 58
Population: as for outcome 50
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 151 | 31
Titers
  hSBA-MenA (PRE): number analyzed (Participants) | 148 | 30
  hSBA-MenA (PRE) | 2 [2 to 2] | 2.2 [1.9 to 2.5]
  hSBA-MenA (PI[M1]): number analyzed (Participants) | 148 | 30
  hSBA-MenA (PI[M1]) | 57.7 [46.1 to 72.1] | 2.3 [1.8 to 2.9]
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 140 | 28
  hSBA-MenA (PI[M12]) | 3.4 [2.8 to 4.1] | 2.1 [1.9 to 2.3]
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 137 | 30
  hSBA-MenA (PI[M24]) | 4.9 [4.0 to 6.0] | 2.3 [2.0 to 2.6]
  hSBA-MenA (PI[M36]): number analyzed (Participants) | 143 | 29
  hSBA-MenA (PI[M36]) | 3.3 [2.8 to 3.9] | 2.1 [1.9 to 2.3]
  hSBA-MenA (PI[M48]): number analyzed (Participants) | 140 | 31
  hSBA-MenA (PI[M48]) | 6 [4.7 to 7.7] | 3.1 [2.3 to 4]
  hSBA-MenC (PRE): number analyzed (Participants) | 146 | 28
  hSBA-MenC (PRE) | 2.1 [2 to 2.2] | 2 [2 to 2]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 151 | 29
  hSBA-MenC (PI[M1]) | 192.5 [160.7 to 230.7] | 45 [23.3 to 86.9]
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 139 | 30
  hSBA-MenC (PI[M12]) | 105.9 [85.6 to 131.1] | 28.6 [14.1 to 58.0]
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 142 | 30
  hSBA-MenC (PI[M24]) | 72.5 [57.3 to 91.6] | 27.1 [12.5 to 58.9]
  hSBA-MenC (PI[M36]): number analyzed (Participants) | 140 | 26
  hSBA-MenC (PI[M36]) | 84.8 [63.7 to 112.9] | 32.4 [15.9 to 66.0]
  hSBA-MenC (PI[M48]): number analyzed (Participants) | 147 | 31
  hSBA-MenC (PI[M48]) | 51.4 [36.9 to 71.7] | 32.4 [14.8 to 71.1]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 141 | 27
  hSBA-MenW-135 (PRE) | 2.1 [2 to 2.2] | 2.1 [1.9 to 2.3]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 119 | 28
  hSBA-MenW-135 (PI[M1]) | 41.7 [30.4 to 57.3] | 2.1 [1.9 to 2.3]
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 121 | 28
  hSBA-MenW-135 (PI[M12]) | 227.9 [176.9 to 293.6] | 2.3 [1.7 to 3.1]
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 134 | 30
  hSBA-MenW-135 (PI[M24]) | 116.5 [92.3 to 147.0] | 3.7 [2.2 to 6.4]
  hSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 139 | 28
  hSBA-MenW-135 (PI[M36]) | 44.5 [33.3 to 59.4] | 2.8 [1.7 to 4.7]
  hSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 143 | 31
  hSBA-MenW-135 (PI[M48]) | 48.3 [36.2 to 64.4] | 2.8 [1.9 to 4.2]
  hSBA-MenY (PRE): number analyzed (Participants) | 127 | 26
  hSBA-MenY (PRE) | 2.1 [2 to 2.2] | 2.1 [1.9 to 2.3]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 139 | 28
  hSBA-MenY (PI[M1]) | 22.5 [16.3 to 31.1] | 2.6 [1.7 to 4.1]
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 150 | 31
  hSBA-MenY (PI[M12]) | 108.8 [84.6 to 140.0] | 3.8 [2.2 to 6.6]
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 132 | 26
  hSBA-MenY (PI[M24]) | 76.3 [57.8 to 100.8] | 6.6 [3.4 to 12.9]
  hSBA-MenY (PI[M36]): number analyzed (Participants) | 133 | 27
  hSBA-MenY (PI[M36]) | 43.0 [30.6 to 60.4] | 5.9 [2.8 to 12.4]
  hSBA-MenY (PI[M48]): number analyzed (Participants) | 129 | 26
  hSBA-MenY (PI[M48]) | 42.1 [30.6 to 58.1] | 13.5 [5.6 to 32.3]

60. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8. This analysis was performed by the GSK Biologicals' laboratory, on the ATP cohort for persistence Year 5.
Time Frame: as for outcome 58
Population: The analysis was performed on subjects from 1 to 2 years of age from the ATP cohort for persistence Year 5, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 5 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 49 | 11
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 41 | 8
  rSBA-MenA (PRE) | 17 | 5
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 49 | 9
  rSBA-MenA (PI[M1]) | 49 | 3
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 48 | 6
  rSBA-MenA (PI[M12]) | 48 | 1
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 48 | 8
  rSBA-MenA (PI[M24]) | 48 | 7
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 45 | 9
  rSBA-MenA (PI[M36]) | 45 | 9
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 40 | 7
  rSBA-MenA (PI[M48]) | 40 | 7
  rSBA-MenC (PRE): number analyzed (Participants) | 45 | 10
  rSBA-MenC (PRE) | 15 | 3
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 48 | 11
  rSBA-MenC (PI[M1]) | 48 | 11
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 47 | 10
  rSBA-MenC (PI[M12]) | 47 | 10
  rSBA-MenC (PI[M24]) | 49 | 11
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 46 | 10
  rSBA-MenC (PI[M36]) | 46 | 10
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 43 | 10
  rSBA-MenC (PI[M48]) | 43 | 9
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 45 | 11
  rSBA-MenW-135 (PRE) | 14 | 3
  rSBA-MenW-135 (PI[M1]) | 49 | 3
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 48 | 10
  rSBA-MenW-135 (PI[M12]) | 48 | 7
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 49 | 8
  rSBA-MenW-135 (PI[M24]) | 48 | 4
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 46 | 8
  rSBA-MenW-135 (PI[M36]) | 45 | 5
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 40 | 9
  rSBA-MenW-135 (PI[M48]) | 37 | 5
  rSBA-MenY (PRE): number analyzed (Participants) | 48 | 10
  rSBA-MenY (PRE) | 30 | 8
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 49 | 10
  rSBA-MenY (PI[M1]) | 49 | 8
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 48 | 10
  rSBA-MenY (PI[M12]) | 48 | 8
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 48 | 11
  rSBA-MenY (PI[M24]) | 48 | 10
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 47 | 9
  rSBA-MenY (PI[M36]) | 47 | 8
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 40 | 10
  rSBA-MenY (PI[M48]) | 39 | 8

61. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs). This analysis was performed by the GSK Biologicals' laboratory, on the ATP cohort for persistence Year 5.
Time Frame: as for outcome 58
Population: as for outcome 60
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 49 | 11
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 41 | 8
  rSBA-MenA (PRE) | 22.6 [11.4 to 44.4] | 45.7 [7.3 to 287.7]
  rSBA-MenA (PI[M1]): number analyzed (Participants) | 49 | 9
  rSBA-MenA (PI[M1]) | 4931.9 [4071.9 to 5973.6] | 16.7 [3.1 to 89.8]
  rSBA-MenA (PI[M12]): number analyzed (Participants) | 48 | 6
  rSBA-MenA (PI[M12]) | 1224.2 [958.4 to 1563.8] | 7.8 [1.4 to 43.7]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 48 | 8
  rSBA-MenA (PI[M24]) | 668.3 [511.6 to 873] | 119.5 [34.5 to 414.8]
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 45 | 9
  rSBA-MenA (PI[M36]) | 578.5 [445.8 to 750.7] | 210.8 [128.8 to 345.2]
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 40 | 7
  rSBA-MenA (PI[M48]) | 782.4 [551.3 to 1110.2] | 392 [192.7 to 797.6]
  rSBA-MenC (PRE): number analyzed (Participants) | 45 | 10
  rSBA-MenC (PRE) | 10.7 [6.7 to 17.1] | 9.4 [3.2 to 27.9]
  rSBA-MenC (PI[M1]): number analyzed (Participants) | 48 | 11
  rSBA-MenC (PI[M1]) | 1115.3 [878.3 to 1416.3] | 536.8 [278.6 to 1034.1]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 47 | 10
  rSBA-MenC (PI[M12]) | 352.4 [251.3 to 494.2] | 249.3 [128.8 to 482.4]
  rSBA-MenC (PI[M24]) | 229.5 [169 to 311.6] | 215.6 [77.6 to 599]
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 46 | 10
  rSBA-MenC (PI[M36]) | 472.4 [285.2 to 782.3] | 229.5 [82 to 642.1]
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 43 | 10
  rSBA-MenC (PI[M48]) | 729.9 [468.4 to 1137.4] | 332 [61.2 to 1802]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 45 | 11
  rSBA-MenW-135 (PRE) | 12.8 [7.4 to 22.2] | 8.4 [3.1 to 22.7]
  rSBA-MenW-135 (PI[M1]) | 6805 [5432.2 to 8524.7] | 12.2 [3.4 to 43.8]
  rSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 48 | 10
  rSBA-MenW-135 (PI[M12]) | 956.5 [710.1 to 1288.3] | 49.4 [13 to 188]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 49 | 8
  rSBA-MenW-135 (PI[M24]) | 408.5 [287.2 to 581.1] | 25.9 [4.5 to 148.3]
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 46 | 8
  rSBA-MenW-135 (PI[M36]) | 486 [316.5 to 746.5] | 52.9 [8.2 to 342.5]
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 40 | 9
  rSBA-MenW-135 (PI[M48]) | 419 [235.1 to 746.7] | 31.3 [5.8 to 167.9]
  rSBA-MenY (PRE): number analyzed (Participants) | 48 | 10
  rSBA-MenY (PRE) | 43.7 [24.5 to 78] | 99.6 [23 to 431]
  rSBA-MenY (PI[M1]): number analyzed (Participants) | 49 | 10
  rSBA-MenY (PI[M1]) | 3555.6 [2928.3 to 4317.3] | 138.7 [29.8 to 645.6]
  rSBA-MenY (PI[M12]): number analyzed (Participants) | 48 | 10
  rSBA-MenY (PI[M12]) | 976.8 [716.8 to 1331.2] | 148 [30.5 to 717.9]
  rSBA-MenY (PI[M24]): number analyzed (Participants) | 48 | 11
  rSBA-MenY (PI[M24]) | 703 [500.8 to 986.9] | 185.1 [59.5 to 576.3]
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 47 | 9
  rSBA-MenY (PI[M36]) | 684 [468.3 to 998.9] | 242.2 [45.3 to 1294.5]
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 40 | 10
  rSBA-MenY (PI[M48]) | 601.5 [365.1 to 991] | 189 [35.8 to 998.1]

62. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: as for outcome 60
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)], Persistence Year 3 [PI(M36)], Persistence Year 4 [PI(M48)]
Population: The analysis was performed on subjects of 2 years and above from the ATP cohort for persistence Year 5, which included all evaluable subjects who had received the vaccine during the vaccination stage and had available assay results for at least one tested antigen at the Year 5 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 98 | 13
Participants
  rSBA-MenA (PRE): number analyzed (Participants) | 81 | 10
  rSBA-MenA (PRE) | 57 | 4
  rSBA-MenA (PI[M1]) | 98 | 13
  rSBA-MenA (PI[M12]) | 98 | 12
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 97 | 12
  rSBA-MenA (PI[M24]) | 97 | 11
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 95 | 13
  rSBA-MenA (PI[M36]) | 95 | 12
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenA (PI[M48]) | 97 | 11
  rSBA-MenC (PRE): number analyzed (Participants) | 94 | 13
  rSBA-MenC (PRE) | 65 | 12
  rSBA-MenC (PI[M1]) | 98 | 13
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 97 | 12
  rSBA-MenC (PI[M12]) | 97 | 12
  rSBA-MenC (PI[M24]) | 98 | 13
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 96 | 13
  rSBA-MenC (PI[M36]) | 96 | 13
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenC (PI[M48]) | 97 | 13
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 86 | 12
  rSBA-MenW-135 (PRE) | 55 | 10
  rSBA-MenW-135 (PI[M1]) | 98 | 13
  rSBA-MenW-135 (PI[M12]) | 98 | 13
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 98 | 12
  rSBA-MenW-135 (PI[M24]) | 98 | 10
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 98 | 12
  rSBA-MenW-135 (PI[M36]) | 98 | 10
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenW-135 (PI[M48]) | 97 | 11
  rSBA-MenY (PRE): number analyzed (Participants) | 94 | 13
  rSBA-MenY (PRE) | 62 | 6
  rSBA-MenY (PI[M1]) | 98 | 13
  rSBA-MenY (PI[M12]) | 98 | 12
  rSBA-MenY (PI[M24]) | 98 | 11
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 97 | 13
  rSBA-MenY (PI[M36]) | 97 | 11
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenY (PI[M48]) | 97 | 11

63. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 61
Time Frame: as for outcome 53
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 98 | 13
Titers
  rSBA-MenA (PRE): number analyzed (Participants) | 81 | 10
  rSBA-MenA (PRE) | 64.3 [41.9 to 98.7] | 35.7 [4.6 to 277.8]
  rSBA-MenA (PI[M1]) | 9195.5 [8097.2 to 10442.6] | 2319 [1337.7 to 4019.9]
  rSBA-MenA (PI[M12]) | 3031.2 [2569.8 to 3575.5] | 491 [157.4 to 1531.1]
  rSBA-MenA (PI[M24]): number analyzed (Participants) | 97 | 12
  rSBA-MenA (PI[M24]) | 1641.7 [1375.5 to 1959.3] | 187.9 [61.2 to 576.6]
  rSBA-MenA (PI[M36]): number analyzed (Participants) | 95 | 13
  rSBA-MenA (PI[M36]) | 1318.4 [1124.3 to 1545.9] | 219.9 [87 to 555.5]
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenA (PI[M48]) | 2365 [1957.2 to 2857.7] | 135.4 [37.6 to 487.1]
  rSBA-MenC (PRE): number analyzed (Participants) | 94 | 13
  rSBA-MenC (PRE) | 44.7 [30.2 to 66.2] | 114 [41.5 to 313.6]
  rSBA-MenC (PI[M1]) | 3604.6 [2921.3 to 4447.7] | 2361.1 [1010.1 to 5518.9]
  rSBA-MenC (PI[M12]): number analyzed (Participants) | 97 | 12
  rSBA-MenC (PI[M12]) | 777.4 [633.7 to 953.7] | 1002 [520 to 1931]
  rSBA-MenC (PI[M24]) | 502.5 [402 to 628.1] | 627.1 [248.2 to 1584.1]
  rSBA-MenC (PI[M36]): number analyzed (Participants) | 96 | 13
  rSBA-MenC (PI[M36]) | 514.4 [409.4 to 646.4] | 865.2 [475.5 to 1574]
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenC (PI[M48]) | 495.2 [386.7 to 634.1] | 742.7 [356.7 to 1546.6]
  rSBA-MenW-135 (PRE): number analyzed (Participants) | 86 | 12
  rSBA-MenW-135 (PRE) | 50.5 [32.4 to 78.8] | 86.8 [29.7 to 253.8]
  rSBA-MenW-135 (PI[M1]) | 13562 [11976.3 to 15357.6] | 2601 [1301.1 to 5199.6]
  rSBA-MenW-135 (PI[M12]) | 3794.4 [3232 to 4454.6] | 462.2 [235.5 to 907.5]
  rSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 98 | 12
  rSBA-MenW-135 (PI[M24]) | 1637.9 [1385.7 to 1936] | 137.4 [42.5 to 443.9]
  rSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 98 | 12
  rSBA-MenW-135 (PI[M36]) | 2098.3 [1783.7 to 2468.3] | 96.6 [28.5 to 327.6]
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenW-135 (PI[M48]) | 2178.4 [1843.2 to 2574.4] | 100.6 [37.9 to 267]
  rSBA-MenY (PRE): number analyzed (Participants) | 94 | 13
  rSBA-MenY (PRE) | 54.3 [35.4 to 83.2] | 15.7 [5.5 to 44.7]
  rSBA-MenY (PI[M1]) | 7167.2 [6324.9 to 8121.8] | 2085.3 [1028.6 to 4227.2]
  rSBA-MenY (PI[M12]) | 2502.4 [2125.3 to 2946.3] | 322.7 [113.1 to 920.9]
  rSBA-MenY (PI[M24]) | 1907.1 [1574.2 to 2310.4] | 112.3 [32 to 394]
  rSBA-MenY (PI[M36]): number analyzed (Participants) | 97 | 13
  rSBA-MenY (PI[M36]) | 1670.6 [1413.6 to 1974.3] | 92.2 [31.9 to 266.4]
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenY (PI[M48]) | 1736 [1430.4 to 2106.8] | 83.3 [29.3 to 236.3]

64. Secondary Outcome: Number of Subjects With rSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: as for outcome 55
Time Frame: Prior to (PRE), one month post vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)], Persistence Year 3 [PI(M36)], Persistence Year 4 [PI(M48)] and Persistence Year 5 [PI(M60)]
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1-2 Years of Age Group
Number analyzed (Participants) | 49 | 11
Participants
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenA (PI[M48]) | 29 | 0
  rSBA-MenA (PI[M60]) | 36 | 0
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenC (PI[M48]) | 44 | 8
  rSBA-MenC (PI[M60]) | 38 | 7
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenW-135 (PI[M48]) | 27 | 0
  rSBA-MenW-135 (PI[M60]) | 17 | 2
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenY (PI[M48]) | 28 | 3
  rSBA-MenY (PI[M60]) | 21 | 2

65. Secondary Outcome: rSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).This analysis was performed by the Health Protection Agency (HPA) laboratory.
Time Frame: as for outcome 64
Population: as for outcome 60
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 49 | 11
Titers
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenA (PI[M48]) | 35.1 [19.4 to 63.4] | 4 [4 to 4]
  rSBA-MenA (PI[M60]) | 37.4 [22.1 to 63.2] | 4 [4 to 4]
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenC (PI[M48]) | 109.7 [62.7 to 192] | 137.2 [22.6 to 831.8]
  rSBA-MenC (PI[M60]) | 48.9 [28.5 to 84] | 26.5 [6.5 to 107.2]
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenW-135 (PI[M48]) | 50.8 [24 to 107.6] | 4 [4 to 4]
  rSBA-MenW-135 (PI[M60]) | 18.2 [9.3 to 35.3] | 7.1 [2.6 to 19.1]
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 45 | 10
  rSBA-MenY (PI[M48]) | 44.9 [22.6 to 89.3] | 12.1 [2.3 to 63.5]
  rSBA-MenY (PI[M60]) | 20.6 [10.9 to 39.2] | 11.7 [2.3 to 59.7]

66. Secondary Outcome: Number of Subjects With rSBA Antibody Titers ≥ the Cut-off Value
Description: as for outcome 55
Time Frame: as for outcome 64
Population: as for outcome 62
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 98 | 13
Participants
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenA (PI[M48]) | 86 | 1
  rSBA-MenA (PI[M60]) | 89 | 2
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenC (PI[M48]) | 96 | 12
  rSBA-MenC (PI[M60]) | 89 | 13
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 96 | 13
  rSBA-MenW-135 (PI[M48]) | 92 | 2
  rSBA-MenW-135 (PI[M60]) | 77 | 0
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 96 | 13
  rSBA-MenY (PI[M48]) | 85 | 1
  rSBA-MenY (PI[M60]) | 77 | 1

67. Secondary Outcome: rSBA Antibody Titers
Description: as for outcome 54
Time Frame: Prior to (PRE), one month after vaccination [PI(M1)], at Persistence Year 1 [PI(M12)], Persistence Year 2 [PI(M24)], Persistence Year 3 [PI(M36)], Persistence Year 4 [PI(M48)] and at Persistence Year 5 [PI(M60)]
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 2- 11 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 98 | 13
Titers
  rSBA-MenA (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenA (PI[M48]) | 123.5 [85.4 to 178.6] | 5 [3.1 to 7.9]
  rSBA-MenA (PI[M60]) | 141.3 [98.2 to 203.4] | 4.7 [3.7 to 6]
  rSBA-MenC (PI[M48]): number analyzed (Participants) | 97 | 13
  rSBA-MenC (PI[M48]) | 118.3 [86 to 162.8] | 206.8 [71.7 to 596.7]
  rSBA-MenC (PI[M60]) | 79.7 [56 to 113.3] | 128 [56.4 to 290.7]
  rSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 96 | 13
  rSBA-MenW-135 (PI[M48]) | 1031.4 [731 to 1455.4] | 8.4 [2.8 to 25.7]
  rSBA-MenW-135 (PI[M60]) | 208.5 [127.9 to 340] | 4 [4 to 4]
  rSBA-MenY (PI[M48]): number analyzed (Participants) | 96 | 13
  rSBA-MenY (PI[M48]) | 216.8 [147.3 to 319.1] | 4.2 [3.8 to 4.7]
  rSBA-MenY (PI[M60]) | 143.3 [88 to 233.4] | 5.5 [2.7 to 11.1]

68. Secondary Outcome: Number of Subjects With hSBA Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: as for outcome 64
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 49 | 11
Participants
  hSBA-MenA (PRE): number analyzed (Participants) | 47 | 11
  hSBA-MenA (PRE) | 0 | 0
  hSBA-MenA (PI[M1]) | 48 | 0
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 47 | 8
  hSBA-MenA (PI[M12]) | 12 | 0
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 43 | 11
  hSBA-MenA (PI[M24]) | 21 | 0
  hSBA-MenA (PI[M36]): number analyzed (Participants) | 46 | 10
  hSBA-MenA (PI[M36]) | 15 | 1
  hSBA-MenA (PI[M48]): number analyzed (Participants) | 44 | 10
  hSBA-MenA (PI[M48]) | 23 | 2
  hSBA-MenA (PI[M60]): number analyzed (Participants) | 45 | 11
  hSBA-MenA (PI[M60]) | 16 | 3
  hSBA-MenC (PRE): number analyzed (Participants) | 45 | 10
  hSBA-MenC (PRE) | 0 | 0
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 48 | 11
  hSBA-MenC (PI[M1]) | 48 | 9
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 46 | 11
  hSBA-MenC (PI[M12]) | 45 | 5
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 45 | 10
  hSBA-MenC (PI[M24]) | 43 | 7
  hSBA-MenC (PI[M36]): number analyzed (Participants) | 46 | 8
  hSBA-MenC (PI[M36]) | 46 | 7
  hSBA-MenC (PI[M48]): number analyzed (Participants) | 45 | 10
  hSBA-MenC (PI[M48]) | 44 | 7
  hSBA-MenC (PI[M60]): number analyzed (Participants) | 48 | 11
  hSBA-MenC (PI[M60]) | 45 | 10
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 44 | 9
  hSBA-MenW-135 (PRE) | 1 | 1
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 41 | 11
  hSBA-MenW-135 (PI[M1]) | 37 | 0
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 42 | 10
  hSBA-MenW-135 (PI[M12]) | 41 | 0
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 42 | 11
  hSBA-MenW-135 (PI[M24]) | 40 | 1
  hSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 45 | 9
  hSBA-MenW-135 (PI[M36]) | 39 | 0
  hSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 45 | 10
  hSBA-MenW-135 (PI[M48]) | 38 | 0
  hSBA-MenW-135 (PI[M60]): number analyzed (Participants) | 46 | 9
  hSBA-MenW-135 (PI[M60]) | 38 | 2
  hSBA-MenY (PRE): number analyzed (Participants) | 45 | 8
  hSBA-MenY (PRE) | 2 | 2
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 48 | 10
  hSBA-MenY (PI[M1]) | 40 | 0
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 48 | 11
  hSBA-MenY (PI[M12]) | 47 | 1
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 41 | 10
  hSBA-MenY (PI[M24]) | 38 | 4
  hSBA-MenY (PI[M36]): number analyzed (Participants) | 43 | 10
  hSBA-MenY (PI[M36]) | 33 | 4
  hSBA-MenY (PI[M48]): number analyzed (Participants) | 41 | 10
  hSBA-MenY (PI[M48]) | 36 | 4
  hSBA-MenY (PI[M60]): number analyzed (Participants) | 45 | 10
  hSBA-MenY (PI[M60]) | 36 | 4

69. Secondary Outcome: hSBA Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: as for outcome 64
Population: as for outcome 60
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group
Number analyzed (Participants) | 49 | 11
Titers
  hSBA-MenA (PRE): number analyzed (Participants) | 47 | 11
  hSBA-MenA (PRE) | 2 [2 to 2] | 2 [2 to 2]
  hSBA-MenA (PI[M1]) | 78.5 [55.7 to 110.4] | 2 [2 to 2]
  hSBA-MenA (PI[M12]): number analyzed (Participants) | 47 | 8
  hSBA-MenA (PI[M12]) | 4.1 [2.8 to 6.1] | 2 [2 to 2]
  hSBA-MenA (PI[M24]): number analyzed (Participants) | 43 | 11
  hSBA-MenA (PI[M24]) | 6.7 [4.3 to 10.3] | 2 [2 to 2]
  hSBA-MenA (PI[M36]): number analyzed (Participants) | 46 | 10
  hSBA-MenA (PI[M36]) | 4.4 [3 to 6.3] | 2.3 [1.7 to 3.3]
  hSBA-MenA (PI[M48]): number analyzed (Participants) | 44 | 10
  hSBA-MenA (PI[M48]) | 8.8 [5.4 to 14.2] | 2.9 [1.6 to 5.3]
  hSBA-MenA (PI[M60]): number analyzed (Participants) | 45 | 11
  hSBA-MenA (PI[M60]) | 5.2 [3.4 to 7.8] | 3.6 [1.8 to 7.2]
  hSBA-MenC (PRE): number analyzed (Participants) | 45 | 10
  hSBA-MenC (PRE) | 2 [2 to 2] | 2 [2 to 2]
  hSBA-MenC (PI[M1]): number analyzed (Participants) | 48 | 11
  hSBA-MenC (PI[M1]) | 252 [193.2 to 328.6] | 38.7 [10.5 to 142.9]
  hSBA-MenC (PI[M12]): number analyzed (Participants) | 46 | 11
  hSBA-MenC (PI[M12]) | 180.1 [121 to 268] | 10.8 [2.5 to 47.7]
  hSBA-MenC (PI[M24]): number analyzed (Participants) | 45 | 10
  hSBA-MenC (PI[M24]) | 137.9 [85.3 to 223] | 33.4 [4.3 to 259.5]
  hSBA-MenC (PI[M36]): number analyzed (Participants) | 46 | 8
  hSBA-MenC (PI[M36]) | 337.9 [215.9 to 528.7] | 57.9 [14.8 to 226.4]
  hSBA-MenC (PI[M48]): number analyzed (Participants) | 45 | 10
  hSBA-MenC (PI[M48]) | 370.2 [214.1 to 640] | 91.9 [9.8 to 858.9]
  hSBA-MenC (PI[M60]): number analyzed (Participants) | 48 | 11
  hSBA-MenC (PI[M60]) | 216.5 [123.6 to 379.1] | 108.7 [21.2 to 557.2]
  hSBA-MenW-135 (PRE): number analyzed (Participants) | 44 | 9
  hSBA-MenW-135 (PRE) | 2.2 [1.8 to 2.5] | 2.3 [1.6 to 3.3]
  hSBA-MenW-135 (PI[M1]): number analyzed (Participants) | 41 | 11
  hSBA-MenW-135 (PI[M1]) | 81.3 [45.4 to 145.7] | 2 [2 to 2]
  hSBA-MenW-135 (PI[M12]): number analyzed (Participants) | 42 | 10
  hSBA-MenW-135 (PI[M12]) | 300.5 [191.2 to 472.1] | 2 [2 to 2]
  hSBA-MenW-135 (PI[M24]): number analyzed (Participants) | 42 | 11
  hSBA-MenW-135 (PI[M24]) | 168.2 [101.8 to 277.8] | 3.1 [1.2 to 8.1]
  hSBA-MenW-135 (PI[M36]): number analyzed (Participants) | 45 | 9
  hSBA-MenW-135 (PI[M36]) | 70.2 [41.4 to 119.1] | 2 [2 to 2]
  hSBA-MenW-135 (PI[M48]): number analyzed (Participants) | 45 | 10
  hSBA-MenW-135 (PI[M48]) | 76.9 [44 to 134.5] | 2 [2 to 2]
  hSBA-MenW-135 (PI[M60]): number analyzed (Participants) | 46 | 9
  hSBA-MenW-135 (PI[M60]) | 59.7 [35.1 to 101.4] | 5.1 [1.2 to 20.9]
  hSBA-MenY (PRE): number analyzed (Participants) | 45 | 8
  hSBA-MenY (PRE) | 2.1 [1.9 to 2.4] | 2.6 [1.7 to 3.8]
  hSBA-MenY (PI[M1]): number analyzed (Participants) | 48 | 10
  hSBA-MenY (PI[M1]) | 46.1 [27.4 to 77.5] | 2 [2 to 2]
  hSBA-MenY (PI[M12]): number analyzed (Participants) | 48 | 11
  hSBA-MenY (PI[M12]) | 160 [107.7 to 237.7] | 3 [1.2 to 7]
  hSBA-MenY (PI[M24]): number analyzed (Participants) | 41 | 10
  hSBA-MenY (PI[M24]) | 121.9 [72 to 206.4] | 8.7 [2.2 to 34.2]
  hSBA-MenY (PI[M36]): number analyzed (Participants) | 43 | 10
  hSBA-MenY (PI[M36]) | 53.9 [28.2 to 102.8] | 7.1 [2 to 25]
  hSBA-MenY (PI[M48]): number analyzed (Participants) | 41 | 10
  hSBA-MenY (PI[M48]) | 74.6 [44.5 to 125.3] | 10 [2.2 to 46.1]
  hSBA-MenY (PI[M60]): number analyzed (Participants) | 45 | 10
  hSBA-MenY (PI[M60]) | 70.6 [38.7 to 128.8] | 11.6 [2.2 to 59.4]

70. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) (1 - < 2 years of age and 2 - < 6 years of age groups) and 50 mm (6 - < 11 years of age groups) of injection site, respectively.
Time Frame: During the 4-day (Day 0-3) follow-up period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available for the vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix 2-6 Years of Age Group: Subjects from 2 to 6 years of age who received one dose of Nimenrix™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
- Nimenrix 6- 11 Years of Age Group: Subjects from 6 to 11 years of age who received one dose of Nimenrix™ vaccine administrated IM by injection in the non-dominant deltoid or the thigh region.
- Mencevax 2- 6 Years of Age Group: Subjects from 2 to 6 years of age who received one dose Mencevax™ vaccine administrated subcutaneous by injection in the non-dominant upper arm.
- Mencevax 6- 11 Years of Age Group: Subjects from 6 to 11 years of age who received one dose of Mencevax™ vaccine administrated subcutaneous by injection in the non-dominant upper arm.
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-6 Years of Age Group | Nimenrix 6- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 6 Years of Age Group | Mencevax 6- 11 Years of Age Group
Number analyzed (Participants) | 228 | 113 | 117 | 73 | 39 | 39
Participants
  Any Pain | 76 | 51 | 84 | 20 | 39 | 39
  Grade 3 Pain | 3 | 2 | 7 | 0 | 1 | 1
  Any Redness | 84 | 44 | 53 | 24 | 8 | 15
  Grade 3 Redness | 8 | 12 | 19 | 1 | 0 | 0
  Any Swelling | 36 | 29 | 42 | 11 | 3 | 6
  Grade 3 Swelling | 3 | 9 | 14 | 0 | 0 | 0

71. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as rectal temperature equal to or above 38.0 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-6 Years of Age Group | Nimenrix 6- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 6 Years of Age Group | Mencevax 6- 11 Years of Age Group
Number analyzed (Participants) | 228 | 113 | 117 | 73 | 39 | 39
Participants
  Any Drowsiness | 63 | 30 | 45 | 25 | 5 | 8
  Grade 3 Drowsiness | 2 | 0 | 1 | 0 | 0 | 0
  Related Drowsiness | 61 | 29 | 45 | 25 | 5 | 8
  Any Fever | 36 | 7 | 11 | 9 | 2 | 1
  Grade 3 Fever >40.0˚C | 2 | 0 | 0 | 0 | 0 | 0
  Related Fever | 32 | 7 | 11 | 9 | 2 | 0
  Any Irritability | 88 | 18 | 23 | 29 | 11 | 5
  Grade 3 Irritability | 2 | 0 | 3 | 0 | 0 | 1
  Related Irritability | 85 | 18 | 21 | 29 | 10 | 4
  Any Loss of appetite | 54 | 16 | 31 | 17 | 6 | 6
  Grade 3 Loss of appetite | 2 | 0 | 1 | 0 | 0 | 0
  Related Loss of appetite | 52 | 16 | 29 | 17 | 5 | 5

72. Secondary Outcome: Number of Subjects With Rash
Description: Rash assessed included hives, idiopathic thrombocytopenic purpura and petechiae.
Time Frame: From administration of the vaccine dose until 6 months later
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 229 | 75 | 231 | 78
Participants | 10 | 6 | 9 | 1

73. Secondary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From administration of the vaccine dose until 6 months later
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 229 | 75 | 231 | 78
Participants | 1 | 0 | 2 | 4

74. Secondary Outcome: Number of Subjects With Adverse Events (AEs) Resulting in an Emergency Room (ER) Visit
Description: Among AEs prompting emergency room visits were: infections, injuries, skin diseases and respiratory diseases.
Time Frame: From administration of the vaccine dose until 6 months later
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 229 | 75 | 231 | 78
Participants | 21 | 8 | 15 | 5

75. Secondary Outcome: Number of Subjects With Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 229 | 75 | 231 | 78
Participants | 121 | 38 | 83 | 24

76. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to 6 Months after vaccination
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Meningitec 1- 2 Years of Age Group | Nimenrix 2- 11 Years of Age Primary Phase Group | Mencevax 2- 11 Years of Age Primary Phase Group
Number analyzed (Participants) | 229 | 75 | 231 | 78
Participants | 5 | 7 | 2 | 1

77. Secondary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 76
Time Frame: From 6 Months after vaccination up to Year 1
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 222 | 221 | 71 | 78
Participants | 0 | 0 | 0 | 0

78. Secondary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 76
Time Frame: From 6 Months after vaccination up to Year 2
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 208 | 215 | 53 | 61
Participants | 0 | 0 | 0 | 0

79. Secondary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 76
Time Frame: From 6 Months following vaccination up to Year 3
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 185 | 201 | 38 | 38
Participants | 0 | 0 | 0 | 0

80. Secondary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 76
Time Frame: From 6 Months following vaccination up to Year 4
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 165 | 192 | 34 | 32
Participants | 0 | 0 | 0 | 0

81. Secondary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 76
Time Frame: From 6 Months following vaccination up to Year 5
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2- 11 Years of Age Group | Meningitec 1- 2 Years of Age Group | Mencevax 2- 11 Years of Age Group
Number analyzed (Participants) | 52 | 99 | 12 | 13
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Day 0-3) follow-up vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Day 0 up to Month 60).
Description: The solicited local and general symptoms were only collected for those subjects with their symptom sheets filled in.
Arm/Group | Nimenrix 1-2 Years of Age Group | Nimenrix 2-11 Years of Age Group | Meningitec 1-2 Years of Age Group | Mencevax 2-11 Years of Age Group
All-Cause Mortality (participants affected / at risk) | 0/229 | 0/231 | 0/75 | 0/78
Serious Adverse Events (participants affected / at risk) | 5/229 | 2/231 | 7/75 | 1/78
Other Adverse Events (participants affected / at risk) | 193/229 | 192/231 | 64/75 | 67/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix 1-2 Years of Age Group (N=229) | Nimenrix 2-11 Years of Age Group (N=231) | Meningitec 1-2 Years of Age Group (N=75) | Mencevax 2-11 Years of Age Group (N=78)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix 1-2 Years of Age Group (N=229) | Nimenrix 2-11 Years of Age Group (N=231) | Meningitec 1-2 Years of Age Group (N=75) | Mencevax 2-11 Years of Age Group (N=78)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 5 | 5 | 3
Pain (General disorders) | 76/228 | 135/230 | 20/73 | 60
Redness (General disorders) | 84/228 | 97/230 | 24/73 | 23
Swelling (General disorders) | 36/228 | 71/230 | 11/73 | 9
Drowsiness (General disorders) | 63/228 | 30/230 | 25/73 | 5
Fever (Rectally) (General disorders) | 36/228 | 18/230 | 9/73 | 3
Irritability (General disorders) | 88/228 | 18/230 | 29/73 | 11
Loss of appetite (General disorders) | 54/228 | 16/230 | 17/73 | 6
Fatigue (General disorders) | 0/228 | 45/117 | 0/73 | 8/39
Gastrointestinal (General disorders) | 0/228 | 23/117 | 0/73 | 5/39
Headache (General disorders) | 0/228 | 31/117 | 0 | 6/39
Pyrexia (General disorders) | 15 | 12 | 10 | 2
Diarrhea (Gastrointestinal disorders) | 11 | 5 | 7 | 1
Teething (Gastrointestinal disorders) | 5 | 0 | 4 | 0
Otitis media (Infections and infestations) | 16 | 12 | 9 | 1
Rhinitis (Infections and infestations) | 19 | 9 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 10 | 8 | 4
Gastroenteritis (Infections and infestations) | 12 | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.